CLINICAL TRIAL: NCT02889796
Title: A Randomized, Double-blind, Placebo- and Active-controlled, Multicenter, Phase 3 Study to Assess the Efficacy and Safety of Filgotinib Administered for 52 Weeks in Combination With Methotrexate to Subjects With Moderately to Severely Active Rheumatoid Arthritis Who Have an Inadequate Response to Methotrexate
Brief Title: Filgotinib in Combination With Methotrexate in Adults With Moderately to Severely Active Rheumatoid Arthritis Who Have an Inadequate Response to Methotrexate
Acronym: FINCH 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Collaborators: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-417-0301; 2016-000568-41 (EudraCT Number)
Record Dates: First submitted 2016-08-31; First posted 2016-09-07 (Estimated); Results first posted 2021-01-19 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — GLPG0634; Adalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Filgotinib 200 mg (Experimental): Filgotinib 200 mg + placebo to match filgotinib 100 mg + placebo to match adalimumab 40 mg in addition to a stable dose of methotrexate (MTX)
  Interventions: Drug: Filgotinib; Drug: Placebo to match filgotinib; Drug: Placebo to match adalimumab; Drug: MTX
- Filgotinib 100 mg (Experimental): Filgotinib 100 mg + placebo to match filgotinib 200 mg + placebo to match adalimumab 40 mg in addition to a stable dose of MTX
  Interventions: Drug: Filgotinib; Drug: Placebo to match filgotinib; Drug: Placebo to match adalimumab; Drug: MTX
- Adalimumab (Active Comparator): Placebo to match filgotinib 200 mg + placebo to match filgotinib 100 mg + adalimumab 40 mg in addition to a stable dose of MTX
  Interventions: Drug: Placebo to match filgotinib; Drug: Adalimumab; Drug: MTX
- Placebo to Filgotinib 200 mg (Experimental): Placebo to match filgotinib 200 mg + placebo to match filgotinib 100 mg + placebo to match adalimumab 40 mg in addition to a stable dose of MTX for up to 24 weeks. After 24 weeks, participants will be rerandomized to filgotinib 200 mg to receive filgotinib 200 mg + placebo to match filgotinib 100 mg + placebo to match adalimumab 40 mg in addition to a stable dose of MTX.
  Interventions: Drug: Filgotinib; Drug: Placebo to match filgotinib; Drug: Placebo to match adalimumab; Drug: MTX
- Placebo to Filgotinib 100 mg (Experimental): Placebo to match filgotinib 200 mg + placebo to match filgotinib 100 mg + placebo to match adalimumab 40 mg in addition to a stable dose of MTX for up to 24 weeks. After 24 weeks, participants will be rerandomized to filgotinib 100 mg to receive filgotinib 100 mg + placebo to match filgotinib 200 mg + placebo to match adalimumab 40 mg in addition to a stable dose of MTX.
  Interventions: Drug: Filgotinib; Drug: Placebo to match filgotinib; Drug: Placebo to match adalimumab; Drug: MTX
- Placebo Never Received Filgotinib (Placebo Comparator): Placebo to match filgotinib 200 mg + placebo to match filgotinib 100 mg + placebo to match adalimumab 40 mg in addition to a stable dose of MTX for up to 24 weeks.
  Interventions: Drug: Placebo to match filgotinib; Drug: Placebo to match adalimumab; Drug: MTX

INTERVENTIONS:
Drug: Filgotinib — 200 mg or 100 mg tablet(s) administered orally once daily
  Other Names: GS-6034
  Arms: Filgotinib 100 mg; Filgotinib 200 mg; Placebo to Filgotinib 100 mg; Placebo to Filgotinib 200 mg
Drug: Placebo to match filgotinib — Tablet(s) administered orally once daily
Drug: Adalimumab — 40 mg administered via subcutaneous injection once every two weeks
  Arms: Adalimumab
Drug: Placebo to match adalimumab — Administered via subcutaneous injection once every two weeks
  Arms: Filgotinib 100 mg; Filgotinib 200 mg; Placebo Never Received Filgotinib; Placebo to Filgotinib 100 mg; Placebo to Filgotinib 200 mg
Drug: MTX — Commercially sourced tablet(s) administered orally

SUMMARY:
The primary objective of this study is to evaluate the effects of filgotinib versus placebo for the treatment of signs and symptoms of rheumatoid arthritis (RA) as measured by the percentage of participants achieving an American College of Rheumatology 20% improvement response (ACR20) at Week 12.

ELIGIBILITY:
Key Inclusion Criteria:

* Have a diagnosis of rheumatoid arthritis (RA) [2010 American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) criteria] , and are ACR functional class I-III.
* Have ≥ 6 swollen joints (from a swollen joint count based on 66 joints (SJC66)) and ≥ 6 tender joints (from a tender joint count based on 68 joints (TJC68)) at both screening and Day 1.
* Ongoing treatment with a stable dose of MTX

Key Exclusion Criteria:

* Previous treatment with any janus kinase (JAK) inhibitor

NOTE: Other protocol defined Inclusion/ Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1759 (Actual)
Dates: Start 2016-08-30 (Actual); Primary Completion 2018-07-04 (Actual); Study Completion 2019-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (230):
- United States (48):
  - Huntsville, Alabama
  - Phoenix, Arizona
  - Tucson, Arizona
  - Covina, California
  - Hemet, California
  - La Jolla, California
  - Palm Desert, California
  - Upland, California
  - Victorville, California
  - Whittier, California
  - Clearwater, Florida
  - DeBary, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Miami Lakes, Florida
  - New Port Richey, Florida
  - Orlando, Florida
  - Plantation, Florida
  - Kansas City, Kansas
  - Wichita, Kansas
  - Elizabethtown, Kentucky
  - Lexington, Kentucky
  - Cumberland, Maryland
  - Hagerstown, Maryland
  - Wheaton, Maryland
  - Detroit, Michigan
  - Saint Clair Shores, Michigan
  - Eagan, Minnesota
  - Hattiesburg, Mississippi
  - Tupelo, Mississippi
  - St Louis, Missouri
  - Toms River, New Jersey
  - Albuquerque, New Mexico
  - Salisbury, North Carolina
  - Bethlehem, Pennsylvania
  - Duncansville, Pennsylvania
  - Philadelphia, Pennsylvania
  - Wyomissing, Pennsylvania
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Orangeburg, South Carolina
  - Memphis, Tennessee
  - Beaumont, Texas
  - Corpus Christi, Texas
  - Dallas, Texas
  - Mesquite, Texas
  - San Antonio, Texas
  - Webster, Texas
- Argentina (7):
  - Buenos Aires
  - Caba
  - Mendoza
  - Quilmes
  - San Fernando
  - San Juan
  - San Miguel de Tucumán
- Victoria Park, Western Australia, Australia
- Belgium (3):
  - Brussels
  - Genk
  - Merksem
- Bulgaria (6):
  - Dobrich
  - Haskovo
  - Plovdiv
  - Sofia
  - Varna
  - Vidin
- Trois-Rivières, Quebec, Canada
- Czechia (6):
  - Prague, Prague
  - Brno
  - Ostrava
  - Ostrava-Poruba
  - Prague
  - Uherské Hradiště
- Germany (3):
  - Frankfurt A Main
  - Hamburg
  - Ratingen
- Hong Kong, Hong Kong
- Hungary (5):
  - Kalocsa, Bács-Kiskun county
  - Szentes, Csongrád megye
  - Székesfehérvár, Fejér
  - Budapest
  - Eger
- India (18):
  - Ahmedabad
  - Bangalore
  - Chennai
  - Delhi
  - Gūrgaon
  - Hyderabad
  - Jaipur
  - Kolkata
  - Lucknow
  - Mangalore
  - Nagpur
  - New Delhi
  - Pune
  - Secunderabad
  - Srikakulam
  - Surat
  - Vadodara
  - Visakhapatnam
- Dublin, Ireland
- Israel (3):
  - Haifa
  - Tel Aviv
  - Tel Litwinsky
- Italy (3):
  - Bologna
  - Catania
  - Milan
- Japan (36):
  - Chiba
  - Fukuoka
  - Hiroshima
  - Iizuka-shi
  - Iruma-gun
  - Izumo
  - Kagoshima
  - Katō
  - Kitakyushu-shi
  - Kobe
  - Kumamoto
  - Kurume-shi
  - Kyoto
  - Miyazaki
  - Morioka
  - Nagaoka
  - Nagasaki
  - Nagoya
  - Narashino
  - Nishinomiya
  - Ōita
  - Sanuki-shi
  - Sapporo
  - Sasebo-shi
  - Sayama-shi
  - Shibata
  - Shinjuku-Ku
  - Shizuoka
  - Suita-shi
  - Takaoka
  - Takasaki-shi
  - Tokorozawa
  - Tokyo
  - Tsukuba
  - Wakayama
  - Yokohama
- Mexico (7):
  - Mérida, Yucatán
  - Chihuahua City
  - Distrito Federal
  - Mexico City
  - Mérida
  - Monterrey
  - Morelia
- Leiden, Netherlands
- New Zealand (5):
  - Papatoetoe, Auckland
  - Auckland
  - Hamilton
  - Newtown
  - Timaru
- Poland (14):
  - Wroclaw, Lower Silesian Voivodeship
  - Bialystok
  - Bydgoszcz
  - Bytom
  - Elblag
  - Gdynia
  - Kartuzy
  - Katowice
  - Krakow
  - Nowa Sól
  - Poznan
  - Tomaszów Lubelski
  - Torun
  - Warsaw
- Romania (4):
  - Oradea, Bihor County
  - Bucharest, București
  - Bacau
  - Târgu Mureş
- Russia (10):
  - Barnaul
  - Chelyabinsk
  - Kazan'
  - Kemerovo
  - Moscow
  - Nizhny Novgorod
  - Saint Petersburg
  - Saratov
  - Vladimir
  - Yaroslavl
- Serbia (2):
  - Belgrade
  - Niška Banja
- Slovakia (4):
  - Bratislava
  - Prievidza
  - Rimavská Sobota
  - Topoľčany
- South Africa (3):
  - Cape Town
  - Durban
  - Johannesburg
- South Korea (8):
  - Anyang-si
  - Busan
  - Daegu
  - Daejeon
  - Gwangju
  - Incheon
  - Jeonju
  - Seoul
- Spain (5):
  - A Coruña
  - Málaga
  - Sabadell
  - Santiago de Compostela
  - Valencia
- Taiwan (7):
  - Changhua
  - Kaohsiung City
  - Keelung
  - Taichung
  - Tainan
  - Taipei
  - Taoyuan District
- Thailand (3):
  - Bangkok
  - Chiang Mai
  - Songkhla
- Ukraine (10):
  - Dnipro
  - Kharkiv
  - Kherson
  - Kiev
  - Kyiv
  - Lutsk
  - Lviv
  - Odesa
  - Vinnytsia
  - Zaporizhzhya
- United Kingdom (5):
  - Poole, England
  - Doncaster
  - Edinburgh
  - Newcastle upon Tyne
  - Warrington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Combe B, Kivitz A, Tanaka Y, van der Heijde D, Matzkies F, Bartok B, et al. Efficacy and safety of filgotinib for patients with rheumatoid arthritis with inadequate response to methotrexate: FINCH 1 primary outcome results. Ann Rheum Dis 2019; 78 (supplement 2):A77.
- [Derived] Tanaka Y, Atsumi T, Aletaha D, Schulze-Koops H, Fukada H, Watson C, Takeuchi T. The Uncoupling of Disease Activity from Joint Structural Progression in Patients with Rheumatoid Arthritis Treated with Filgotinib. Rheumatol Ther. 2025 Feb;12(1):53-66. doi: 10.1007/s40744-024-00725-7. Epub 2024 Nov 26. PMID 39592547
- [Derived] Buch MH, Walker D, Edwards CJ, Barry J, Akroyd L, Ekoka Omoruyi EV, Taylor PC. Efficacy and safety of filgotinib in patients with moderately active rheumatoid arthritis and an inadequate response to methotrexate. Rheumatology (Oxford). 2025 Apr 1;64(4):1661-1671. doi: 10.1093/rheumatology/keae486. PMID 39331638
- [Derived] Taylor PC, Downie B, Han L, Hawtin R, Hertz A, Moots RJ, Takeuchi T. Patients with High Baseline Neutrophil-to-Lymphocyte Ratio Exhibit Better Response to Filgotinib as Treatment for Rheumatoid Arthritis. Rheumatol Ther. 2024 Oct;11(5):1383-1392. doi: 10.1007/s40744-024-00695-w. Epub 2024 Jul 10. PMID 38985247
- [Derived] Curtis JR, Emery P, Downie B, Zhong Y, Liu J, Han L, Hawtin RE, Burmester GR. Filgotinib Demonstrates Efficacy in Rheumatoid Arthritis Independent of Smoking Status: Post Hoc Analysis of Phase 3 Trials and Claims-Based Analysis. Rheumatol Ther. 2024 Feb;11(1):177-189. doi: 10.1007/s40744-023-00619-0. Epub 2023 Dec 6. PMID 38057656
- [Derived] Balsa A, Wassenberg S, Tanaka Y, Tournadre A, Orzechowski HD, Rajendran V, Lendl U, Stiers PJ, Watson C, Caporali R, Galloway J, Verschueren P. Effect of Filgotinib on Body Mass Index (BMI) and Effect of Baseline BMI on the Efficacy and Safety of Filgotinib in Rheumatoid Arthritis. Rheumatol Ther. 2023 Dec;10(6):1555-1574. doi: 10.1007/s40744-023-00599-1. Epub 2023 Sep 25. PMID 37747626
- [Derived] Tanaka Y, Taylor PC, Elboudwarej E, Hertz A, Shao X, Malkov VA, Matsushima H, Emoto K, Downie B, Takeuchi T. Filgotinib Modulates Inflammation-Associated Peripheral Blood Protein Biomarkers in Adults with Active Rheumatoid Arthritis and Prior Inadequate Response to Methotrexate. Rheumatol Ther. 2023 Oct;10(5):1335-1348. doi: 10.1007/s40744-023-00583-9. Epub 2023 Jul 25. PMID 37490202
- [Derived] Tanaka Y, Atsumi T, Aletaha D, Bartok B, Pechonkina A, Han L, Emoto K, Kano S, Rajendran V, Takeuchi T. Benefit of Filgotinib, a JAK1 Preferential Inhibitor, in Rheumatoid Arthritis Patients with Previous Rapid Radiographic Progression: Post Hoc Analysis of Two Trials. Rheumatol Ther. 2023 Feb;10(1):161-185. doi: 10.1007/s40744-022-00503-3. Epub 2022 Nov 3. PMID 36327094
- [Derived] Combe B, Besuyen R, Gomez-Centeno A, Matsubara T, Sancho Jimenez JJ, Yin Z, Buch MH. Geographic Analysis of the Safety and Efficacy of Filgotinib in Rheumatoid Arthritis. Rheumatol Ther. 2023 Feb;10(1):35-51. doi: 10.1007/s40744-022-00494-1. Epub 2022 Oct 7. PMID 36205910
- [Derived] Bingham CO 3rd, Walker D, Nash P, Lee SJ, Ye L, Hu H, Khalid JM, Combe B. The impact of filgotinib on patient-reported outcomes and health-related quality of life for patients with active rheumatoid arthritis: a post hoc analysis of Phase 3 studies. Arthritis Res Ther. 2022 Jan 3;24(1):11. doi: 10.1186/s13075-021-02677-7. PMID 34980223
- [Derived] Combe B, Kivitz A, Tanaka Y, van der Heijde D, Simon JA, Baraf HSB, Kumar U, Matzkies F, Bartok B, Ye L, Guo Y, Tasset C, Sundy JS, Jahreis A, Genovese MC, Mozaffarian N, Landewe RBM, Bae SC, Keystone EC, Nash P. Filgotinib versus placebo or adalimumab in patients with rheumatoid arthritis and inadequate response to methotrexate: a phase III randomised clinical trial. Ann Rheum Dis. 2021 Jul;80(7):848-858. doi: 10.1136/annrheumdis-2020-219214. Epub 2021 Jan 27. PMID 33504485

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Asia, South Africa, Australia, Europe, North America, South America, and New Zealand. The first participant was screened on 30 August 2016. The last study visit occurred on 20 June 2019.
Pre-assignment Details: 2582 participants were screened.
Groups:
- Filgotinib 200 mg: Participants were administered a filgotinib 200 mg tablet orally, once daily + placebo to match (PTM) filgotinib 100 mg tablet orally, once daily + PTM adalimumab 40 mg subcutaneous (SC) injection, once every 2 weeks in addition to a weekly stable dose of MTX, orally for median exposure of up to 52.1 weeks.
- Filgotinib 100 mg: Participants were administered a filgotinib 100 mg tablet orally, once daily + PTM filgotinib 200 mg tablet orally, once daily + PTM adalimumab 40 mg SC injection, once every 2 weeks in addition to a weekly stable dose of MTX, orally for median exposure of up to 52.1 weeks.
- Adalimumab: Participants were administered PTM filgotinib 200 mg tablet orally, once daily + PTM filgotinib 100 mg tablet orally, once daily + adalimumab 40 mg SC injection, once every 2 weeks in addition to a weekly stable dose of MTX, orally for median exposure of up to 52.1 weeks.
- Placebo to Filgotinib 200 mg: Participants in the placebo arm were administered a PTM filgotinib 200 mg tablet orally, once daily+ a PTM filgotinib 100 mg tablet orally, once daily + PTM adalimumab 40 mg SC injection, once every 2 weeks in addition to a weekly stable dose of MTX, orally for median exposure of up to 24 weeks. Then the participants in the placebo arm were rerandomized to filgotinib 200 mg and were administered a filgotinib 200 mg tablet orally, once daily + PTM filgotinib 100 mg tablet orally, once daily + PTM adalimumab 40 mg SC injection, once every 2 weeks in addition to a weekly stable dose of MTX, orally for median exposure of up to 28.1 weeks.
- Placebo to Filgotinib 100 mg: Participants in the placebo arm were administered a PTM filgotinib 200 mg tablet orally, once daily+ a PTM filgotinib 100 mg tablet orally, once daily + PTM adalimumab 40 mg SC injection, once every 2 weeks in addition to a weekly stable dose of MTX, orally for median exposure of up to 24 weeks. Then the participants in the placebo arm were rerandomized to filgotinib 100 mg and were administered a filgotinib 100 mg tablet orally, once daily + PTM filgotinib 200 mg tablet orally, once daily + PTM adalimumab 40 mg SC injection, once every 2 weeks in addition to a weekly stable dose of MTX, orally for median exposure of up to 28.1 weeks.
- Placebo Never Received Filgotinib: Participants in the placebo arm were administered a PTM filgotinib 200 mg tablet orally, once daily+ a PTM filgotinib 100 mg tablet orally, once daily + PTM adalimumab 40 mg SC injection, once every 2 weeks in addition to a weekly stable dose of MTX, orally for median exposure of up to 24 weeks.
Period: Overall Study
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo to Filgotinib 200 mg | Placebo to Filgotinib 100 mg | Placebo Never Received Filgotinib
Started | 477 | 480 | 325 | 190 | 191 | 96
Completed | 424 | 422 | 281 | 181 | 185 | 24 (Completed 24 weeks of placebo treatment and not rerandomized to Filgotinib 200 mg or 100 mg groups)
Not Completed | 53 | 58 | 44 | 9 | 6 | 72
Not completed — Withdrew Consent | 18 | 29 | 20 | 1 | 2 | 35
Not completed — Investigator's Discretion | 10 | 9 | 10 | 3 | 0 | 15
Not completed — Adverse Event | 17 | 8 | 8 | 4 | 1 | 7
Not completed — Lost to Follow-up | 5 | 7 | 2 | 0 | 2 | 6
Not completed — Protocol Violation | 0 | 1 | 3 | 0 | 0 | 4
Not completed — Non-compliance With Study Drug | 0 | 2 | 0 | 0 | 1 | 2
Not completed — Death | 1 | 1 | 0 | 1 | 0 | 1
Not completed — Pregnancy | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Randomized but not Dosed | 2 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who received at least 1 dose of study drug.
Groups:
- Placebo: The Placebo arm includes all participants who received placebo in the study. Participants were administered a PTM filgotinib 200 mg tablet orally, once daily+ a PTM filgotinib 100 mg tablet orally, once daily + PTM adalimumab 40 mg SC injection, once every 2 weeks in addition to a weekly stable dose of MTX, orally for median exposure of up to 24 weeks. Participants could be rerandomized to filgotinib 200 mg or 100 mg groups.
- Total: Total of all reporting groups
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo | Total
Number analyzed (Participants) | 475 | 480 | 325 | 475 | 1755
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (12.8) | 53 (12.6) | 53 (12.9) | 53 (12.8) | 53 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 379 | 399 | 266 | 391 | 1435
  Male | 96 | 81 | 59 | 84 | 320
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not Permitted=local regulators did not allow collection of race information.
  Participants
    Race: American Indian or Alaska Native | 27 | 27 | 20 | 29 | 103
    Race: Asian: Japanese | 40 | 41 | 28 | 38 | 147
    Race: Asian: Chinese/Taiwanese/Hong Kong Chinese | 13 | 12 | 8 | 18 | 51
    Race: Asian: Korean | 13 | 10 | 4 | 7 | 34
    Race: Asian: Other | 56 | 52 | 25 | 46 | 179
    Race: Black or African American | 6 | 7 | 10 | 12 | 35
    Race: Native Hawaiian or Pacific Islander | 1 | 0 | 0 | 2 | 3
    Race: White | 312 | 324 | 229 | 319 | 1184
    Race: Other | 7 | 6 | 1 | 3 | 17
    Race: Not Permitted | 0 | 1 | 0 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not Permitted=local regulators did not allow collection of ethnicity information.
  Participants
    Ethnicity: Hispanic or Latino | 67 | 71 | 54 | 70 | 262
    Ethnicity: Not Hispanic or Latino | 404 | 399 | 268 | 400 | 1471
    Ethnicity: Not Permitted | 4 | 10 | 3 | 5 | 22
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 47 | 55 | 37 | 60 | 199
  South Africa | 12 | 11 | 3 | 8 | 34
  South Korea | 12 | 10 | 4 | 7 | 33
  Spain | 14 | 3 | 6 | 7 | 30
  Germany | 5 | 6 | 5 | 4 | 20
  New Zealand | 5 | 5 | 3 | 5 | 18
  United Kingdom | 1 | 2 | 4 | 6 | 13
  Canada | 4 | 4 | 3 | 1 | 12
  Israel | 4 | 1 | 2 | 4 | 11
  Belgium | 2 | 3 | 4 | 1 | 10
  Italy | 2 | 1 | 2 | 1 | 6
  Netherlands | 0 | 1 | 0 | 1 | 2
  Australia | 0 | 1 | 0 | 0 | 1
  Ireland | 0 | 1 | 0 | 0 | 1
  Poland | 78 | 82 | 64 | 74 | 298
  Ukraine | 66 | 73 | 41 | 55 | 235
  India | 40 | 39 | 19 | 39 | 137
  Russia | 34 | 32 | 22 | 30 | 118
  Hungary | 12 | 12 | 5 | 17 | 46
  Bulgaria | 7 | 7 | 6 | 14 | 34
  Czechia | 7 | 7 | 7 | 13 | 34
  Romania | 12 | 6 | 2 | 11 | 31
  Serbia | 1 | 7 | 8 | 5 | 21
  Slovakia | 2 | 2 | 1 | 3 | 8
  Mexico | 33 | 33 | 25 | 34 | 125
  Argentina | 15 | 17 | 10 | 15 | 57
  Taiwan | 12 | 9 | 7 | 16 | 44
  Thailand | 7 | 6 | 6 | 4 | 23
  Hong Kong | 1 | 3 | 1 | 2 | 7
  Japan | 40 | 41 | 28 | 38 | 147

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved an American College of Rheumatology (ACR) 20% Improvement (ACR20) Response at Week 12
Description: ACR20 response is achieved when the participant has: ≥20% improvement (reduction) from baseline in tender joint count based on 68 joints (TJC68), swollen joint count based on 66 joints (SJC66) and in at least 3 of the following 5 items: physician's global assessment of disease activity (PGA) and subject's global assessment of disease activity (SGA) assessed using visual analog scale (VAS) on a scale of 0-100 (0 and 100 indicating no disease activity and maximum disease activity)participant's pain assessment using VAS on a scale of 0-100 (0 and 100 indicating no pain and unbearable pain) health assessment questionnaire-disability index (HAQ-DI) score contains 20 questions,8 components: dressing/ grooming, arising, eating, walking, hygiene, reach, grip and activities and scored on a scale of 0-3 (0 and 3 indicating without difficulty and unable to do); high-sensitivity C-reactive protein (hsCRP). Participants with missing outcomes were set as non-responders.
Time Frame: Week 12
Population: The Full Analysis Set included participants who were randomized and received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Filgotinib 200 mg: Participants were administered a filgotinib 200 mg tablet orally, once daily + placebo to match (PTM) filgotinib 100 mg tablet orally, once daily + PTM adalimumab 40 mg subcutaneous (SC) injection, once every 2 weeks in addition to a weekly stable dose of methotrexate (MTX), orally for median exposure of up to 52.1 weeks.
- Adalimumab: Participants were administered a PTM filgotinib 200 mg tablet orally, once daily + PTM filgotinib 100 mg tablet orally, once daily + adalimumab 40 mg SC injection, once every 2 weeks in addition to a weekly stable dose of MTX, orally for median exposure of up to 52.1 weeks.
- Placebo: The Placebo arm included all participants who received placebo in the study. Participants were administered a PTM filgotinib 200 mg tablet orally, once daily+ a PTM filgotinib 100 mg tablet orally, once daily + PTM adalimumab 40 mg SC injection, once every 2 weeks in addition to a weekly stable dose of MTX, orally for median exposure of 24 weeks. Participants could be rerandomized to filgotinib 200 mg or 100 mg groups.
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo
Number analyzed (Participants) | 475 | 480 | 325 | 475
percentage of participants | 76.6 [72.7 to 80.5] | 69.8 [65.6 to 74.0] | 70.5 [65.3 to 75.6] | 49.9 [45.3 to 54.5]
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; Filgotinib 200 mg vs Placebo at Week 12; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 26.7, 95% CI 2-sided [20.6 to 32.8]
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; Filgotinib 100 mg vs Placebo at Week 12; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 19.9, 95% CI 2-sided [13.6 to 26.2]

2. Secondary Outcome: Change From Baseline in the Health Assessment Questionnaire-Disability Index (HAQ-DI) Score at Week 12
Description: The HAQ-DI score is defined as the average of the scores of eight functional categories (dressing and grooming, arising, eating, walking, hygiene, reach, grip, and other activities), usually completed by the participant. Responses in each functional category are collected as 0 (without any difficulty) to 3 (unable to do a task in that area), with or without aids or devices. The eight category scores are averaged into an overall HAQ-DI score on a scale from 0 (no disability) to 3 (completely disabled). When 6 or more categories are non-missing, total possible score is 3. If more than 2 categories are missing, the HAQ-DI score is set to missing. Negative change from baseline indicates improvement (less disability).
Time Frame: Baseline; Week 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Filgotinib 200 mg: Participants were administered a filgotinib 200 mg tablet orally, once daily + a placebo to match (PTM) filgotinib 100 mg tablet orally, once daily + PTM adalimumab 40 mg subcutaneous (SC) injection, once every 2 weeks in addition to a weekly stable dose of MTX, orally for median exposure of up to 52.1 weeks.
- Filgotinib 100 mg: Participants were administered a filgotinib 100 mg tablet orally, once daily + a PTM filgotinib 200 mg tablet orally, once daily + PTM adalimumab 40 mg SC injection, once every 2 weeks in addition to a weekly stable dose of MTX, orally for median exposure of up to 52.1 weeks
- Adalimumab: Participants were administered a PTM filgotinib 200 mg tablet orally, once daily + a PTM filgotinib 100 mg tablet orally, once daily + adalimumab 40 mg SC injection, once every 2 weeks in addition to a weekly stable dose of MTX, orally for median exposure of up to 52.1 weeks.
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo
Number analyzed (Participants) | 475 | 480 | 325 | 475
score on a scale
  Baseline | 1.59 (0.611) | 1.55 (0.625) | 1.59 (0.600) | 1.63 (0.613)
  Change from Baseline at Week 12: number analyzed (Participants) | 457 | 459 | 311 | 435
  Change from Baseline at Week 12 | -0.69 (0.613) | -0.56 (0.564) | -0.61 (0.560) | -0.42 (0.544)
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; Filgotinib 200 mg vs Placebo at Week 12. LS-Mean, 95% CI, and P-value were provided from mixed effects model for repeated measures (MMRM). Missing change scores were not imputed using the MMRM approach assuming an unstructured variance-covariance matrix for the repeated measures; Test type: Superiority; p < 0.001, Mixed effects model for repeated measure — MMRM model included treatment, visit, treatment by visit, stratification factors, and baseline value as fixed effects, and participants being the random effect; Least Squares Mean Difference = -0.29, 95% CI 2-sided [-0.36 to -0.22], Standard Error of Mean 0.034
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; Filgotinib 100 mg vs Placebo at Week 12. LS-Mean, 95% CI, and P-value were provided from MMRM. Missing change scores were not imputed using the MMRM approach assuming an unstructured variance-covariance matrix for the repeated measures; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.17, 95% CI 2-sided [-0.24 to -0.10], Standard Error of Mean 0.034

3. Secondary Outcome: Percentage of Participants Who Achieved Disease Activity Score for 28 Joint Count Using C-Reactive Protein [DAS28 (CRP)] < 2.6 at Week 12
Description: The DAS28 score is a measure of the participant's disease activity calculated using the tender joint counts (28 joints), swollen joint counts (28 joints), SGA (VAS: 0 = no disease activity to 100 = maximum disease activity), and hsCRP (CRP = hsCRP) for a total possible score of 1 to 9.4. Higher values indicate higher disease activity. Participants with missing outcomes were set as non-responders.
Time Frame: Week 12
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo
Number analyzed (Participants) | 475 | 480 | 325 | 475
percentage of participants | 34.1 [29.7 to 38.5] | 23.8 [19.8 to 27.7] | 23.7 [18.9 to 28.5] | 9.3 [6.6 to 12.0]
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; Filgotinib 200 mg vs Placebo at Week 12; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 24.8, 95% CI 2-sided [19.6 to 30.0]
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; Filgotinib 100 mg vs Placebo at Week 12; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 14.5, 95% CI 2-sided [9.7 to 19.3]
Statistical Analysis 3: Comparison: Filgotinib 200 mg vs Adalimumab; Filgotinib 200 mg vs Adalimumab at Week 12; Test type: Non-Inferiority — For non-inferiority test, the approach proposed by Liu 2014 was used to demonstrate that each filgotinib dose preserves more than 50% of the effect of adalimumab on the response rate of DAS28 (CRP) < 2.6 using non-responder imputation (NRI); p < 0.001, Method proposed by [Liu 2014] — P-value of non-inferiority test was calculated from approach proposed by [Liu 2014]
Statistical Analysis 4: Comparison: Filgotinib 100 mg vs Adalimumab; Filgotinib 100 mg vs Adalimumab at Week 12; Test type: Non-Inferiority — For non-inferiority test, the approach proposed by Liu 2014 was used to demonstrate that each filgotinib dose preserves more than 50% of the effect of adalimumab on the response rate of DAS28 (CRP) < 2.6 using NRI; p = 0.002, Method proposed by [Liu 2014] — P-value of non-inferiority test was calculated from approach proposed by [Liu 2014]
Statistical Analysis 5: Comparison: Filgotinib 200 mg vs Adalimumab; Filgotinib 200 mg vs Adalimumab at Week 12; Test type: Superiority; p = 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 10.4, 95% CI 2-sided [3.9 to 17.0]
Statistical Analysis 6: Comparison: Filgotinib 100 mg vs Adalimumab; Filgotinib 100 mg vs Adalimumab at Week 12; Test type: Superiority; p = 0.99, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 0.1, 95% CI 2-sided [-6.2 to 6.3]

4. Secondary Outcome: Change From Baseline in Modified Total Sharp Score (mTSS) at Week 24
Description: Participant's radiographs of bilateral hands, wrists and feet are taken and evaluated through central review using the mTSS method. The mTSS (range [0-448]) is defined as the erosion score (range [0-280]) plus the joint space narrowing (JSN) score (range [0-168]). An erosion score of 0 to 5 is given to each joint in the hands and wrists, and a score of 0 to 10 is given to each joint in the feet where 0 indicates no erosion while 5 or 10 indicates extensive loss of bone (maximum erosion). JSN is scored from 0 to 4, with 0 indicating normal or no narrowing and 4 indicating complete loss of joint space. The maximal TSS is 448. Negative change in value indicates improvement (less erosion of bone, normal joint spaces).
Time Frame: Baseline; Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo: The Placebo arm included all participants who received placebo in the study. Participants were administered a PTM filgotinib 200 mg tablet orally, once daily+ a PTM filgotinib 100 mg tablet orally, once daily + PTM adalimumab 40 mg SC injection, once every 2 weeks in addition to a weekly stable dose of MTX, orally for median exposure of up to 24 weeks. Participants could be rerandomized to filgotinib 200 mg or filgotinib 100 mg.
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo
Number analyzed (Participants) | 467 | 471 | 319 | 466
score on a scale
  Baseline | 32.47 (47.939) | 36.70 (53.065) | 34.82 (55.013) | 31.60 (53.217)
  Change from Baseline at Week 24: number analyzed (Participants) | 405 | 404 | 271 | 351
  Change from Baseline at Week 24 | 0.13 (0.937) | 0.17 (0.905) | 0.16 (0.948) | 0.37 (1.417)
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; Filgotinib 200 mg vs Placebo at Week 24. LS-Mean, 95% CI, and P-value were provided from MMRM. Missing change scores were not imputed using the MMRM approach assuming an unstructured variance-covariance matrix for the repeated measures; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.27, 95% CI 2-sided [-0.43 to -0.12], Standard Error of Mean 0.078
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; Filgotinib 100 mg vs Placebo at Week 24. LS-Mean, 95% CI, and P-value were provided from MMRM. Missing change scores were not imputed using the MMRM approach assuming an unstructured variance-covariance matrix for the repeated measures; Test type: Superiority; p = 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.25, 95% CI 2-sided [-0.40 to -0.10], Standard Error of Mean 0.078

5. Secondary Outcome: Percentage of Participants Who Achieved DAS28 (CRP) ≤ 3.2 at Week 12
Description: The DAS28 score is a measure of the participant's disease activity calculated using the tender joint counts (28 joints), swollen joint counts (28 joints), SGA (VAS: 0 = no disease activity to 100 = maximum disease activity), and hsCRP for a total possible score of 1 to 9.4. Higher values indicate higher disease activity. Participants with missing outcomes were set as non-responders.
Time Frame: Week 12
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo
Number analyzed (Participants) | 475 | 480 | 325 | 475
percentage of participants | 49.7 [45.1 to 54.3] | 38.8 [34.3 to 43.2] | 43.4 [37.8 to 48.9] | 23.4 [19.5 to 27.3]
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; Filgotinib 200 mg vs Placebo at Week 12; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 26.3, 95% CI 2-sided [20.2 to 32.4]
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; Filgotinib 100 mg vs Placebo at Week 12; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 15.4, 95% CI 2-sided [9.4 to 21.4]
Statistical Analysis 3: Comparison: Filgotinib 200 mg vs Adalimumab; Filgotinib 200 mg vs Adalimumab at Week 12; Test type: Non-Inferiority — For non-inferiority test, the approach proposed by Liu 2014 was used to demonstrate that each filgotinib dose preserves more than 50% of the effect of adalimumab on the response rate of DAS28 (CRP) ≤ 3.2 using NRI; p < 0.001, Method proposed by [Liu 2014] — P-value of non-inferiority test was calculated from approach proposed by [Liu 2014]
Statistical Analysis 4: Comparison: Filgotinib 100 mg vs Adalimumab; Filgotinib 100 mg vs Adalimumab at Week 12; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 3]; p = 0.054, Method proposed by [Liu 2014] — P-value of non-inferiority test was calculated from approach proposed by [Liu 2014]
Statistical Analysis 5: Comparison: Filgotinib 200 mg vs Adalimumab; Filgotinib 200 mg vs Adalimumab at Week 12; Test type: Superiority; p = 0.069, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 6.3, 95% CI 2-sided [-1.0 to 13.6]
Statistical Analysis 6: Comparison: Filgotinib 100 mg vs Adalimumab; Filgotinib 100 mg vs Adalimumab at Week 12; Test type: Superiority; p = 0.18, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = -4.6, 95% CI 2-sided [-11.8 to 2.6]

6. Secondary Outcome: Change From Baseline in 36-Item Short Form Survey (SF-36) Physical Component Summary (PCS) Score at Week 12
Description: The SF-36 is a 36-item, self-reported, generic, comprehensive, and health-related quality of life questionnaire based on 8 health domains in 2 components: physical well-being (physical functioning, role-physical, bodily pain, general health perceptions), mental well-being (vitality, social functioning, role-emotional, and mental health). Each domain is scored by summing the individual items and transforming the scores into a 0 to 100 scale with highest possible score of 100. Higher scores indicate better health status or functioning. Positive change in value indicates improvement and better quality of life.
Time Frame: Baseline; Week 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo
Number analyzed (Participants) | 473 | 479 | 323 | 474
score on a scale
  Baseline | 33.4 (7.17) | 33.6 (7.75) | 32.8 (7.74) | 32.9 (7.11)
  Change from Baseline at Week 12: number analyzed (Participants) | 459 | 463 | 310 | 440
  Change from Baseline at Week 12 | 9.2 (8.10) | 8.5 (7.72) | 8.4 (7.89) | 5.8 (7.10)
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; Filgotinib 200 mg vs Placebo at Week 12. LS-Mean, 95% CI, and P-value were provided from MMRM. Missing change scores were not imputed using the MMRM approach assuming an unstructured variance-covariance matrix for the repeated measures; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 3.7, 95% CI 2-sided [2.8 to 4.6], Standard Error of Mean 0.47
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 3.1, 95% CI 2-sided [2.2 to 4.0], Standard Error of Mean 0.46

7. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Score at Week 12
Description: FACIT-Fatigue scale is a brief, 13-item, symptom-specific questionnaire that specifically assesses the self-reported severity of fatigue and its impact upon daily activities and functioning in the past 7 days. The FACIT-Fatigue uses 0 (not at all) to 4 (very much) numeric rating scales for a total possible score of 0 to 52. Positive change in value indicates improvement (no or less severity of fatigue).
Time Frame: Baseline; Week 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo
Number analyzed (Participants) | 472 | 477 | 319 | 469
score on a scale
  Baseline | 27.6 (10.68) | 27.8 (10.60) | 27.2 (10.20) | 26.9 (10.34)
  Change from Baseline at Week 12: number analyzed (Participants) | 452 | 455 | 304 | 432
  Change from Baseline at Week 12 | 9.2 (9.82) | 9.1 (10.15) | 8.8 (9.19) | 6.8 (9.89)
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 2.8, 95% CI 2-sided [1.7 to 3.9], Standard Error of Mean 0.56
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 2.6, 95% CI 2-sided [1.5 to 3.7], Standard Error of Mean 0.55

8. Secondary Outcome: Percentage of Participants Who Achieved ACR 50% Improvement (ACR50) at Weeks 2, 4, 12, and 24
Description: ACR50 response is achieved when the participant has: ≥50% improvement (reduction) from baseline in TJC68, SJC66 and in at least 3 of the following 5 items: PGA and SGA assessed using VAS on a scale of 0-100 [0 and 100 indicating no disease activity and maximum disease activity]; subject's pain assessment using VAS on a scale of 0-100 [0 and 100 indicating no pain and unbearable pain]; HAQ-DI score contains 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities and scored on a scale of 0-3 [0 and 3 indicating without difficulty and unable to do]; hsCRP. Participants with missing outcomes were set as non-responders.
Time Frame: Weeks 2, 4, 12, and 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo
Number analyzed (Participants) | 475 | 480 | 325 | 475
percentage of participants
  Week 2 | 9.1 [6.4 to 11.7] | 5.8 [3.6 to 8.0] | 6.8 [3.9 to 9.7] | 1.1 [0.0 to 2.1]
  Week 4 | 22.3 [18.5 to 26.2] | 12.9 [9.8 to 16.0] | 17.2 [13.0 to 21.5] | 5.9 [3.7 to 8.1]
  Week 12 | 47.2 [42.6 to 51.8] | 36.5 [32.0 to 40.9] | 35.1 [29.7 to 40.4] | 19.8 [16.1 to 23.5]
  Week 24 | 57.9 [53.3 to 62.4] | 52.7 [48.1 to 57.3] | 52.3 [46.7 to 57.9] | 33.3 [28.9 to 37.6]
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; Filgotinib 200 mg vs Placebo at Week 2; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 8.0, 95% CI 2-sided [5.1 to 10.9]
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; Filgotinib 100 mg vs Placebo at Week 2; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 4.8, 95% CI 2-sided [2.3 to 7.3]
Statistical Analysis 3: Comparison: Filgotinib 200 mg vs Placebo; Filgotinib 200 mg vs Placebo at Week 4; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 16.4, 95% CI 2-sided [11.9 to 20.9]
Statistical Analysis 4: Comparison: Filgotinib 100 mg vs Placebo; Filgotinib 100 mg vs Placebo at Week 4; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 7.0, 95% CI 2-sided [3.1 to 10.9]
Statistical Analysis 5: Comparison: Filgotinib 200 mg vs Placebo; Filgotinib 200 mg vs Placebo at Week 12; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 27.4, 95% CI 2-sided [21.4 to 33.3]
Statistical Analysis 6: Comparison: Filgotinib 100 mg vs Placebo; Filgotinib 100 mg vs Placebo at Week 12; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 16.7, 95% CI 2-sided [10.9 to 22.5]
Statistical Analysis 7: Comparison: Filgotinib 200 mg vs Placebo; Filgotinib 200 mg vs Placebo at Week 24; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 24.6, 95% CI 2-sided [18.3 to 31.0]
Statistical Analysis 8: Comparison: Filgotinib 100 mg vs Placebo; Filgotinib 100 mg vs Placebo at Week 24; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 19.4, 95% CI 2-sided [13.1 to 25.8]

9. Secondary Outcome: Percentage of Participants Who Achieved ACR50 at Weeks 36, and 52
Description: as for outcome 8
Time Frame: Weeks 36, and 52
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo to Filgotinib 200 mg | Placebo to Filgotinib 100 mg
Number analyzed (Participants) | 475 | 480 | 325 | 190 | 191
percentage of participants
  Week 36 | 63.2 [58.7 to 67.6] | 57.7 [53.2 to 62.2] | 57.5 [52.0 to 63.1] | 67.9 [61.0 to 74.8] | 63.4 [56.3 to 70.4]
  Week 52 | 64.2 [59.8 to 68.6] | 60.6 [56.2 to 65.1] | 62.2 [56.7 to 67.6] | 68.4 [61.5 to 75.3] | 66.0 [59.0 to 72.9]

10. Secondary Outcome: Percentage of Participants Who Achieved ACR 70% Improvement (ACR70) at Weeks 2, 4, 12, and 24
Description: ACR70 response is achieved when the participant has: ≥70% improvement (reduction) from baseline in TJC68, SJC66 and in at least 3 of the following 5 items: PGA and SGA assessed using VAS on a scale of 0-100 [0 and 100 indicating no disease activity and maximum disease activity]; subject's pain assessment using VAS on a scale of 0-100 [0 and 100 indicating no pain and unbearable pain]; HAQ-DI score contains 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities and scored on a scale of 0-3 [0 and 3 indicating without difficulty and unable to do]; hsCRP. Participants with missing outcomes were set as non-responders.
Time Frame: Weeks 2, 4, 12, and 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo
Number analyzed (Participants) | 475 | 480 | 325 | 475
percentage of participants
  Week 2 | 2.7 [1.2 to 4.3] | 1.3 [0.2 to 2.3] | 0.9 [0.0 to 2.1] | 0.4 [0.0 to 1.1]
  Week 4 | 9.1 [6.4 to 11.7] | 3.3 [1.6 to 5.0] | 3.7 [1.5 to 5.9] | 1.5 [0.3 to 2.7]
  Week 12 | 26.1 [22.1 to 30.2] | 18.5 [15.0 to 22.1] | 14.2 [10.2 to 18.1] | 6.7 [4.4 to 9.1]
  Week 24 | 36.2 [31.8 to 40.6] | 29.6 [25.4 to 33.8] | 29.5 [24.4 to 34.7] | 14.9 [11.6 to 18.3]
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; Filgotinib 200 mg vs Placebo at Week 2; Test type: Superiority; p = 0.008, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 2.3, 95% CI 2-sided [0.5 to 4.1]
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; Filgotinib 100 mg vs Placebo at Week 2; Test type: Superiority; p = 0.18, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 0.8, 95% CI 2-sided [-0.5 to 2.2]
Statistical Analysis 3: Comparison: Filgotinib 200 mg vs Placebo; Filgotinib 200 mg vs Placebo at Week 4; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 7.6, 95% CI 2-sided [4.6 to 10.6]
Statistical Analysis 4: Comparison: Filgotinib 100 mg vs Placebo; Filgotinib 100 mg vs Placebo at Week 4; Test type: Superiority; p = 0.067, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 1.9, 95% CI 2-sided [-0.3 to 4.0]
Statistical Analysis 5: Comparison: Filgotinib 200 mg vs Placebo; Filgotinib 200 mg vs Placebo at Week 12; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 19.4, 95% CI 2-sided [14.6 to 24.1]
Statistical Analysis 6: Comparison: Filgotinib 100 mg vs Placebo; Filgotinib 100 mg vs Placebo at Week 12; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 11.8, 95% CI 2-sided [7.5 to 16.2]
Statistical Analysis 7: Comparison: Filgotinib 200 mg vs Placebo; Filgotinib 200 mg vs Placebo at Week 24; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 21.3, 95.0% CI 2-sided [15.7 to 26.9]
Statistical Analysis 8: Comparison: Filgotinib 100 mg vs Placebo; Filgotinib 100 mg vs Placebo at Week 24; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 14.6, 95% CI 2-sided [9.2 to 20.0]

11. Secondary Outcome: Percentage of Participants Who Achieved ACR70 at Weeks 36, and 52
Description: as for outcome 10
Time Frame: Weeks 36, and 52
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo to Filgotinib 200 mg | Placebo to Filgotinib 100 mg
Number analyzed (Participants) | 475 | 480 | 325 | 190 | 191
percentage of participants
  Week 36 | 40.2 [35.7 to 44.7] | 35.4 [31.0 to 39.8] | 32.9 [27.7 to 38.2] | 44.7 [37.4 to 52.1] | 34.6 [27.5 to 41.6]
  Week 52 | 44.4 [39.8 to 49.0] | 39.0 [34.5 to 43.4] | 41.2 [35.7 to 46.7] | 48.4 [41.1 to 55.8] | 37.7 [30.6 to 44.8]

12. Secondary Outcome: Percentage of Participants Who Achieved ACR20 Response at Weeks 2, 4, and 24
Description: ACR20 response is achieved when the participant has: ≥20% improvement (reduction) from baseline in TJC68, SJC66 and in at least 3 of the following 5 items: PGA and SGA assessed using VAS on a scale of 0-100 [0 and 100 indicating no disease activity and maximum disease activity]; subject's pain assessment using VAS on a scale of 0-100 [0 and 100 indicating no pain and unbearable pain]; HAQ-DI score contains 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities and scored on a scale of 0-3 [0 and 3 indicating without difficulty and unable to do]; hsCRP. Participants with missing outcomes were set as non-responders.
Time Frame: Weeks 2, 4, and 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo
Number analyzed (Participants) | 475 | 480 | 325 | 475
percentage of participants
  Week 2 | 37.3 [32.8 to 41.7] | 27.5 [23.4 to 31.6] | 33.5 [28.3 to 38.8] | 14.9 [11.6 to 18.3]
  Week 4 | 51.6 [47.0 to 56.2] | 45.6 [41.1 to 50.2] | 47.1 [41.5 to 52.7] | 31.8 [27.5 to 36.1]
  Week 24 | 78.1 [74.3 to 81.9] | 77.7 [73.9 to 81.5] | 74.5 [69.6 to 79.4] | 59.2 [54.6 to 63.7]
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; Filgotinib 200 mg vs Placebo at Week 2; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 22.3, 95% CI 2-sided [16.7 to 27.9]
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; Filgotinib 100 mg vs Placebo at Week 2; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 12.6, 95% CI 2-sided [7.2 to 17.9]
Statistical Analysis 3: Comparison: Filgotinib 200 mg vs Placebo; Filgotinib 200 mg vs Placebo at Week 4; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 19.8, 95% CI 2-sided [13.4 to 26.1]
Statistical Analysis 4: Comparison: Filgotinib 100 mg vs Placebo; Filgotinib 100 mg vs Placebo at Week 4; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 13.8, 95% CI 2-sided [7.5 to 20.2]
Statistical Analysis 5: Comparison: Filgotinib 200 mg vs Placebo; Filgotinib 200 mg vs Placebo at Week 24; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 18.9, 95% CI 2-sided [13.0 to 24.9]
Statistical Analysis 6: Comparison: Filgotinib 100 mg vs Placebo; Filgotinib 100 mg vs Placebo at Week 24; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 18.6, 95% CI 2-sided [12.6 to 24.5]

13. Secondary Outcome: Percentage of Participants Who Achieved ACR20 Response at Weeks 36, and 52
Description: as for outcome 12
Time Frame: Weeks 36, and 52
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo to Filgotinib 200 mg | Placebo to Filgotinib 100 mg
Number analyzed (Participants) | 475 | 480 | 325 | 190 | 191
percentage of participants
  Week 36 | 82.9 [79.5 to 86.4] | 79.2 [75.4 to 82.9] | 76.3 [71.5 to 81.1] | 90.5 [86.1 to 95.0] | 86.9 [81.9 to 92.0]
  Week 52 | 82.9 [79.5 to 86.4] | 79.6 [75.9 to 83.3] | 77.8 [73.2 to 82.5] | 86.3 [81.2 to 91.5] | 85.9 [80.7 to 91.1]

14. Secondary Outcome: Change From Baseline in Individual ACR Component: HAQ-DI at Weeks 2, 4, and 24
Description: The HAQ-DI score is defined as the average of the scores of eight functional categories (dressing and grooming, arising, eating, walking, hygiene, reach, grip, and other activities), usually completed by the participant. Responses in each functional category are collected as 0 (without any difficulty) to 3 (unable to do a task in that area), with or without aids or devices. The eight category scores are averaged into an overall HAQ-DI score on a scale from 0 (no disability) to 3 (completely disabled). A negative change from baseline indicates improvement.
Time Frame: Baseline; Weeks 2, 4, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo
Number analyzed (Participants) | 475 | 480 | 325 | 475
score on a scale
  Baseline | 1.59 (0.611) | 1.55 (0.625) | 1.59 (0.600) | 1.63 (0.613)
  Change from Baseline at Week 2: number analyzed (Participants) | 463 | 474 | 317 | 466
  Change from Baseline at Week 2 | -0.30 (0.443) | -0.22 (0.406) | -0.29 (0.440) | -0.15 (0.357)
  Change from Baseline at Week 4: number analyzed (Participants) | 469 | 471 | 320 | 461
  Change from Baseline at Week 4 | -0.43 (0.493) | -0.33 (0.454) | -0.40 (0.460) | -0.26 (0.431)
  Change from Baseline at Week 24: number analyzed (Participants) | 418 | 423 | 283 | 376
  Change from Baseline at Week 24 | -0.82 (0.632) | -0.75 (0.597) | -0.78 (0.632) | -0.62 (0.598)
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; Filgotinib 200 mg vs Placebo at Week 2. LS-Mean, 95% CI, and P-value were provided from MMRM. Missing change scores were not imputed using the MMRM approach assuming an unstructured variance-covariance matrix for the repeated measures; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.17, 95% CI 2-sided [-0.22 to -0.12], Standard Error of Mean 0.025
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; Filgotinib 100 mg vs Placebo at Week 2. LS-Mean, 95% CI, and P-value were provided from MMRM. Missing change scores were not imputed using the MMRM approach assuming an unstructured variance-covariance matrix for the repeated measures; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.09, 95% CI 2-sided [-0.14 to -0.04], Standard Error of Mean 0.025
Statistical Analysis 3: Comparison: Filgotinib 200 mg vs Placebo; Filgotinib 200 mg vs Placebo at Week 4. LS-Mean, 95% CI, and P-value were provided from MMRM. Missing change scores were not imputed using the MMRM approach assuming an unstructured variance-covariance matrix for the repeated measures; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.19, 95% CI 2-sided [-0.24 to -0.13], Standard Error of Mean 0.028
Statistical Analysis 4: Comparison: Filgotinib 100 mg vs Placebo; Filgotinib 100 mg vs Placebo at Week 4. LS-Mean, 95% CI, and P-value were provided from MMRM. Missing change scores were not imputed using the MMRM approach assuming an unstructured variance-covariance matrix for the repeated measures; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.10, 95% CI 2-sided [-0.15 to -0.04], Standard Error of Mean 0.028
Statistical Analysis 5: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.27, 95% CI 2-sided [-0.34 to -0.19], Standard Error of Mean 0.037
Statistical Analysis 6: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.19, 95% CI 2-sided [-0.26 to -0.11], Standard Error of Mean 0.037

15. Secondary Outcome: Change From Baseline in Individual ACR Component: HAQ-DI at Weeks 36, and 52
Description: as for outcome 14
Time Frame: Baseline; Weeks 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo to Filgotinib 200 mg | Placebo to Filgotinib 100 mg
Number analyzed (Participants) | 475 | 480 | 325 | 190 | 191
score on a scale
  Baseline | 1.59 (0.611) | 1.55 (0.625) | 1.59 (0.600) | 1.68 (0.578) | 1.58 (0.603)
  Change from Baseline at Week 36: number analyzed (Participants) | 412 | 417 | 275 | 180 | 188
  Change from Baseline at Week 36 | -0.88 (0.633) | -0.80 (0.611) | -0.81 (0.634) | -0.96 (0.637) | -0.69 (0.610)
  Change from Baseline at Week 52: number analyzed (Participants) | 400 | 398 | 265 | 173 | 177
  Change from Baseline at Week 52 | -0.93 (0.649) | -0.85 (0.621) | -0.85 (0.647) | -0.99 (0.644) | -0.73 (0.650)

16. Secondary Outcome: Change From Baseline in Individual ACR Component: Tender Joint Count Based on 68 Joints (TJC68) at Weeks 2, 4, 12, and 24
Description: TJC was examined on 68 joints of the fingers, elbows, hips, knees, ankles, and toes distal for pain in response to pressure or passive motion at the study time points. Joint pain was scored as 0 = Absent; 1 = Present for each joint. The overall Tender Joint Count ranged from 0 to 68. A negative change from baseline indicates improvement.
Time Frame: Baseline; Weeks 2, 4, 12, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: tender joint count
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo
Number analyzed (Participants) | 475 | 480 | 325 | 475
tender joint count
  Baseline | 25 (13.5) | 25 (13.4) | 24 (13.2) | 24 (13.5)
  Change from Baseline at Week 2: number analyzed (Participants) | 464 | 473 | 317 | 464
  Change from Baseline at Week 2 | -8 (10.1) | -7 (9.3) | -7 (8.8) | -5 (9.0)
  Change from Baseline at Week 4: number analyzed (Participants) | 469 | 471 | 320 | 461
  Change from Baseline at Week 4 | -11 (11.1) | -10 (10.3) | -9 (9.2) | -8 (10.5)
  Change from Baseline at Week 12: number analyzed (Participants) | 458 | 458 | 311 | 435
  Change from Baseline at Week 12 | -17 (11.1) | -15 (10.7) | -15 (9.9) | -13 (11.6)
  Change from Baseline at Week 24: number analyzed (Participants) | 418 | 423 | 283 | 375
  Change from Baseline at Week 24 | -20 (12.1) | -19 (10.9) | -18 (11.1) | -17 (11.7)
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 14, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -3, 95% CI 2-sided [-4.0 to -2.0], Standard Error of Mean 0.6
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 14, analysis 2]; Test type: Superiority; p = 0.010, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -2.0, 95% CI 2-sided [-3.0 to -0.0], Standard Error of Mean 0.6
Statistical Analysis 3: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 14, analysis 3]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -3.0, 95% CI 2-sided [-5.0 to -2.0], Standard Error of Mean 0.6
Statistical Analysis 4: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 14, analysis 4]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -2.0, 95% CI 2-sided [-4.0 to -1.0], Standard Error of Mean 0.6
Statistical Analysis 5: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -4.0, 95% CI 2-sided [-5.0 to -2.0], Standard Error of Mean 0.6
Statistical Analysis 6: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -3.0, 95% CI 2-sided [-4.0 to -1.0], Standard Error of Mean 0.6
Statistical Analysis 7: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -3.0, 95% CI 2-sided [-4.0 to -2.0], Standard Error of Mean 0.5
Statistical Analysis 8: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -2.0, 95% CI 2-sided [-3.0 to -1.0], Standard Error of Mean 0.5

17. Secondary Outcome: Change From Baseline in Individual ACR Component: TJC68 at Weeks 36, and 52
Description: as for outcome 16
Time Frame: Baseline; Weeks 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: tender joint count
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo to Filgotinib 200 mg | Placebo to Filgotinib 100 mg
Number analyzed (Participants) | 475 | 480 | 325 | 190 | 191
tender joint count
  Baseline | 25 (13.5) | 25 (13.4) | 24 (13.2) | 25 (12.8) | 24 (12.9)
  Change from Baseline at Week 36: number analyzed (Participants) | 411 | 417 | 275 | 178 | 188
  Change from Baseline at Week 36 | -21 (11.9) | -20 (11.2) | -19 (11.0) | -21 (11.4) | -19 (11.5)
  Change from Baseline at Week 52: number analyzed (Participants) | 400 | 397 | 265 | 173 | 177
  Change from Baseline at Week 52 | -21 (12.2) | -21 (11.4) | -20 (11.4) | -21 (11.9) | -20 (11.2)

18. Secondary Outcome: Change From Baseline in Individual ACR Component: Swollen Joint Count Based on 66 Joints (SJC66) at Weeks 2, 4, 12, and 24
Description: The total SJC66 was based on 66 joints (same 68 joints counted in TJC68 minus hips). It was derived as the sum of all "1s" (presence of a joint swelling was scored as "1" and the absence of swelling was scored as "0," provided the joint was not replaced or could not be assessed due to other reasons) thus collected with no penalty considered for the joints not assessed or those which had been replaced. The range for SJC66 is 0 to 66. A negative change from baseline indicates improvement.
Time Frame: Baseline; Weeks 2, 4, 12, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: swollen joint count
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo
Number analyzed (Participants) | 475 | 480 | 325 | 475
swollen joint count
  Baseline | 15 (8.5) | 15 (8.5) | 16 (8.4) | 16 (8.5)
  Change from Baseline at Week 2: number analyzed (Participants) | 464 | 473 | 317 | 464
  Change from Baseline at Week 2 | -6 (6.7) | -5 (6.8) | -6 (5.8) | -5 (6.9)
  Change from Baseline at Week 4: number analyzed (Participants) | 469 | 471 | 320 | 461
  Change from Baseline at Week 4 | -8 (7.1) | -8 (7.8) | -7 (6.6) | -6 (7.8)
  Change from Baseline at Week 12: number analyzed (Participants) | 458 | 458 | 311 | 435
  Change from Baseline at Week 12 | -11 (7.5) | -11 (8.1) | -11 (7.1) | -10 (8.4)
  Change from Baseline at Week 24: number analyzed (Participants) | 418 | 423 | 283 | 375
  Change from Baseline at Week 24 | -13 (7.8) | -13 (7.4) | -13 (6.9) | -12 (7.7)
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 14, analysis 1]; Test type: Superiority; p = 0.002, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -1.0, 95% CI 2-sided [-2.0 to -0.0], Standard Error of Mean 0.4
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 14, analysis 2]; Test type: Superiority; p = 0.047, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -1.0, 95% CI 2-sided [-2.0 to -0.0], Standard Error of Mean 0.4
Statistical Analysis 3: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 14, analysis 3]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -2.0, 95% CI 2-sided [-3.0 to -1.0], Standard Error of Mean 0.4
Statistical Analysis 4: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 14, analysis 4]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -2.0, 95% CI 2-sided [-3.0 to -1.0], Standard Error of Mean 0.4
Statistical Analysis 5: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -2.0, 95% CI 2-sided [-3.0 to -1.0], Standard Error of Mean 0.4
Statistical Analysis 6: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -2.0, 95% CI 2-sided [-2.0 to -1.0], Standard Error of Mean 0.4
Statistical Analysis 7: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -2.0, 95% CI 2-sided [-3.0 to -1.0], Standard Error of Mean 0.3
Statistical Analysis 8: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -1.0, 95.0% CI 2-sided [-2.0 to -1.0], Standard Error of Mean 0.3

19. Secondary Outcome: Change From Baseline in Individual ACR Component: SJC66 at Weeks 36, and 52
Description: as for outcome 18
Time Frame: Baseline; Weeks 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: swollen joint count
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo to Filgotinib 200 mg | Placebo to Filgotinib 100 mg
Number analyzed (Participants) | 475 | 480 | 325 | 190 | 191
swollen joint count
  Baseline | 15 (8.5) | 15 (8.5) | 16 (8.4) | 16 (8.2) | 15 (7.9)
  Change from Baseline at Week 36: number analyzed (Participants) | 411 | 417 | 275 | 178 | 188
  Change from Baseline at Week 36 | -14 (7.8) | -13 (7.6) | -14 (7.1) | -14 (7.3) | -13 (7.2)
  Change from Baseline at Week 52: number analyzed (Participants) | 400 | 397 | 265 | 173 | 177
  Change from Baseline at Week 52 | -14 (8.1) | -13 (7.6) | -14 (7.5) | -14 (7.8) | -13 (7.4)

20. Secondary Outcome: Change From Baseline in Individual ACR Component: Subject's Global Assessment of Disease Activity (SGA) at Weeks 2, 4, 12, and 24
Description: SGA was assessed by the participant using a VAS on a scale of 0 (no disease activity) to 100 (maximum disease activity). A negative change from baseline indicates improvement.
Time Frame: Baseline; Weeks 2, 4, 12, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo: The Placebo arm included all participants who received placebo in the study. Participants were administered a PTM filgotinib 200 mg tablet orally, once daily+ a PTM filgotinib 100 mg tablet orally, once daily + PTM adalimumab 40 mg SC injection, once every 2 weeks in addition to a weekly stable dose of MTX, orally for median exposure of up to 24 weeks.. Participants could be rerandomized to filgotinib 200 mg or filgotinib 100 mg.
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo
Number analyzed (Participants) | 475 | 480 | 325 | 475
score on a scale
  Baseline | 67 (19.2) | 65 (19.7) | 67 (19.1) | 68 (18.7)
  Change from Baseline at Week 2: number analyzed (Participants) | 464 | 474 | 318 | 466
  Change from Baseline at Week 2 | -16 (20.1) | -11 (18.4) | -13 (18.1) | -8 (17.2)
  Change from Baseline at Week 4: number analyzed (Participants) | 469 | 472 | 319 | 461
  Change from Baseline at Week 4 | -22 (21.5) | -16 (20.8) | -19 (20.8) | -13 (20.2)
  Change from Baseline at Week 12: number analyzed (Participants) | 457 | 458 | 311 | 435
  Change from Baseline at Week 12 | -33 (24.8) | -28 (24.7) | -28 (23.2) | -21 (24.8)
  Change from Baseline at Week 24: number analyzed (Participants) | 418 | 423 | 283 | 376
  Change from Baseline at Week 24 | -39 (25.8) | -36 (24.9) | -36 (24.9) | -31 (26.9)
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 14, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -9.0, 95% CI 2-sided [-11.0 to -7.0], Standard Error of Mean 1.1
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 14, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -5.0, 95% CI 2-sided [-7.0 to -2.0], Standard Error of Mean 1.1
Statistical Analysis 3: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 14, analysis 3]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -9.0, 95% CI 2-sided [-12.0 to -7.0], Standard Error of Mean 1.3
Statistical Analysis 4: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 14, analysis 4]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -5.0, 95% CI 2-sided [-7.0 to -2.0], Standard Error of Mean 1.3
Statistical Analysis 5: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -13.0, 95% CI 2-sided [-16.0 to -10.0], Standard Error of Mean 1.5
Statistical Analysis 6: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -10.0, 95% CI 2-sided [-12.0 to -7.0], Standard Error of Mean 1.5
Statistical Analysis 7: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -11.0, 95% CI 2-sided [-14.0 to -7.0], Standard Error of Mean 1.6
Statistical Analysis 8: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -8.0, 95% CI 2-sided [-11.0 to -5.0], Standard Error of Mean 1.6

21. Secondary Outcome: Change From Baseline in Individual ACR Component: SGA at Weeks 36, and 52
Description: as for outcome 20
Time Frame: Baseline; Weeks 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo to Filgotinib 200 mg | Placebo to Filgotinib 100 mg
Number analyzed (Participants) | 475 | 480 | 325 | 190 | 191
score on a scale
  Baseline | 67 (19.2) | 65 (19.7) | 67 (19.1) | 70 (17.8) | 66 (18.7)
  Change from Baseline at Week 36: number analyzed (Participants) | 412 | 417 | 274 | 180 | 188
  Change from Baseline at Week 36 | -42 (24.2) | -39 (25.3) | -39 (25.2) | -45 (24.7) | -38 (25.5)
  Change from Baseline at Week 52: number analyzed (Participants) | 400 | 398 | 265 | 173 | 177
  Change from Baseline at Week 52 | -44 (24.4) | -41 (25.4) | -42 (25.7) | -45 (27.6) | -41 (25.3)

22. Secondary Outcome: Change From Baseline in Individual ACR Component: Physician's Global Assessment of Disease Activity (PGA) at Weeks 2, 4, 12, and 24
Description: PGA was assessed by the physician using a VAS on a scale of 0 (no disease activity) to 100 (maximum disease activity). A negative change from baseline indicates improvement.
Time Frame: Baseline; Weeks 2, 4, 12, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo: The Placebo arm included all participants who received placebo in the study. Participants were administered a PTM filgotinib 200 mg tablet orally, once daily+ a PTM filgotinib 100 mg tablet orally, once daily + PTM adalimumab 40 mg SC injection, once every 2 weeks in addition to a weekly stable dose of MTX, orally for median exposure of up to 24 weeks. Participants were rerandomized to filgotinib 200 mg or filgotinib 100 mg.
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo
Number analyzed (Participants) | 475 | 480 | 325 | 475
score on a scale
  Baseline | 66 (16.0) | 65 (16.5) | 67 (15.5) | 66 (16.2)
  Change from Baseline at Week 2: number analyzed (Participants) | 463 | 469 | 315 | 463
  Change from Baseline at Week 2 | -20 (19.3) | -18 (18.5) | -19 (17.9) | -13 (17.8)
  Change from Baseline at Week 4: number analyzed (Participants) | 468 | 466 | 318 | 457
  Change from Baseline at Week 4 | -28 (21.2) | -26 (19.7) | -26 (19.6) | -20 (19.6)
  Change from Baseline at Week 12: number analyzed (Participants) | 457 | 450 | 308 | 433
  Change from Baseline at Week 12 | -41 (20.2) | -39 (20.3) | -39 (20.4) | -34 (22.4)
  Change from Baseline at Week 24: number analyzed (Participants) | 413 | 419 | 283 | 373
  Change from Baseline at Week 24 | -48 (19.2) | -46 (19.6) | -47 (19.4) | -42 (20.4)
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 14, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -8.0, 95% CI 2-sided [-10.0 to -6.0], Standard Error of Mean 1.1
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 14, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -6.0, 95% CI 2-sided [-8.0 to -4.0], Standard Error of Mean 1.1
Statistical Analysis 3: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 14, analysis 3]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -8.0, 95% CI 2-sided [-11.0 to -6.0], Standard Error of Mean 1.2
Statistical Analysis 4: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 14, analysis 4]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -7.0, 95% CI 2-sided [-9.0 to -5.0], Standard Error of Mean 1.2
Statistical Analysis 5: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -8.0, 95% CI 2-sided [-10.0 to -6.0], Standard Error of Mean 1.2
Statistical Analysis 6: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -7.0, 95% CI 2-sided [-10.0 to -5.0], Standard Error of Mean 1.2
Statistical Analysis 7: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -8.0, 95% CI 2-sided [-11.0 to -6.0], Standard Error of Mean 1.1
Statistical Analysis 8: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -7.0, 95% CI 2-sided [-10.0 to -5.0], Standard Error of Mean 1.1

23. Secondary Outcome: Change From Baseline in Individual ACR Component: PGA at Weeks 36, and 52
Description: as for outcome 22
Time Frame: Baseline; Weeks 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo to Filgotinib 200 mg | Placebo to Filgotinib 100 mg
Number analyzed (Participants) | 475 | 480 | 325 | 190 | 191
score on a scale
  Baseline | 66 (16.0) | 65 (16.5) | 67 (15.5) | 68 (15.6) | 64 (16.3)
  Change from Baseline at Week 36: number analyzed (Participants) | 409 | 416 | 273 | 176 | 187
  Change from Baseline at Week 36 | -51 (19.0) | -49 (19.8) | -50 (18.6) | -53 (19.5) | -47 (20.0)
  Change from Baseline at Week 52: number analyzed (Participants) | 400 | 398 | 265 | 173 | 177
  Change from Baseline at Week 52 | -53 (18.2) | -50 (19.2) | -52 (18.9) | -54 (19.7) | -50 (19.3)

24. Secondary Outcome: Change From Baseline in Individual ACR Component: Subject's Pain Assessment at Weeks 2, 4, 12, and 24
Description: The participant assessed their pain severity using a VAS on a scale of 0 (no pain) to 100 (severe pain). A negative change from baseline indicates improvement.
Time Frame: Baseline; Weeks 2, 4, 12, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo
Number analyzed (Participants) | 475 | 480 | 325 | 475
score on a scale
  Baseline | 65 (20.4) | 64 (20.1) | 64 (19.5) | 66 (19.0)
  Change from Baseline at Week 2: number analyzed (Participants) | 463 | 474 | 317 | 466
  Change from Baseline at Week 2 | -16 (21.0) | -12 (18.7) | -13 (20.4) | -7 (18.2)
  Change from Baseline at Week 4: number analyzed (Participants) | 469 | 471 | 319 | 461
  Change from Baseline at Week 4 | -21 (23.7) | -18 (20.9) | -18 (21.9) | -12 (20.8)
  Change from Baseline at Week 12: number analyzed (Participants) | 457 | 458 | 311 | 435
  Change from Baseline at Week 12 | -31 (26.9) | -29 (25.3) | -27 (23.6) | -21 (26.0)
  Change from Baseline at Week 24: number analyzed (Participants) | 418 | 423 | 283 | 376
  Change from Baseline at Week 24 | -38 (27.0) | -37 (25.6) | -35 (24.2) | -30 (27.0)
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 14, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -9.0, 95% CI 2-sided [-12.0 to -7.0], Standard Error of Mean 1.2
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 14, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -6.0, 95% CI 2-sided [-8.0 to -3.0], Standard Error of Mean 1.2
Statistical Analysis 3: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 14, analysis 3]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -9.0, 95% CI 2-sided [-12.0 to -7.0], Standard Error of Mean 1.3
Statistical Analysis 4: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 14, analysis 4]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -6.0, 95% CI 2-sided [-9.0 to -4.0], Standard Error of Mean 1.3
Statistical Analysis 5: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -12.0, 95% CI 2-sided [-15.0 to -9.0], Standard Error of Mean 1.5
Statistical Analysis 6: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -10.0, 95% CI 2-sided [-13.0 to -7.0], Standard Error of Mean 1.5
Statistical Analysis 7: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -11.0, 95% CI 2-sided [-14.0 to -7.0], Standard Error of Mean 1.6
Statistical Analysis 8: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -9.0, 95% CI 2-sided [-12.0 to -6.0], Standard Error of Mean 1.6

25. Secondary Outcome: Change From Baseline in Individual ACR Component: Subject's Pain Assessment at Weeks 36, and 52
Description: as for outcome 24
Time Frame: Baseline; Weeks 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo to Filgotinib 200 mg | Placebo to Filgotinib 100 mg
Number analyzed (Participants) | 475 | 480 | 325 | 190 | 191
score on a scale
  Baseline | 65 (20.4) | 64 (20.1) | 64 (19.5) | 68 (18.0) | 65 (19.2)
  Change from Baseline at Week 36: number analyzed (Participants) | 412 | 417 | 274 | 180 | 188
  Change from Baseline at Week 36 | -40 (26.3) | -38 (26.2) | -37 (25.5) | -44 (24.9) | -39 (25.9)
  Change from Baseline at Week 52: number analyzed (Participants) | 400 | 398 | 265 | 173 | 177
  Change from Baseline at Week 52 | -43 (26.2) | -41 (25.9) | -41 (25.6) | -45 (26.6) | -41 (25.6)

26. Secondary Outcome: Change From Baseline in Individual ACR Component: High-Sensitivity C-Reactive Protein (hsCRP) at Weeks 2, 4, 12, and 24
Time Frame: Baseline; Weeks 2, 4, 12, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo
Number analyzed (Participants) | 475 | 480 | 325 | 475
mg/L
  Baseline | 16.13 (21.005) | 16.74 (22.982) | 14.56 (18.003) | 16.25 (24.051)
  Change from Baseline at Week 2: number analyzed (Participants) | 455 | 467 | 315 | 463
  Change from Baseline at Week 2 | -10.85 (20.154) | -7.67 (17.888) | -8.03 (15.594) | -0.07 (17.244)
  Change from Baseline at Week 4: number analyzed (Participants) | 465 | 468 | 319 | 456
  Change from Baseline at Week 4 | -9.99 (21.146) | -8.44 (20.201) | -7.17 (16.896) | -1.12 (19.940)
  Change from Baseline at Week 12: number analyzed (Participants) | 456 | 454 | 308 | 431
  Change from Baseline at Week 12 | -11.00 (18.659) | -9.55 (21.330) | -7.85 (20.632) | -3.26 (22.711)
  Change from Baseline at Week 24: number analyzed (Participants) | 416 | 419 | 281 | 370
  Change from Baseline at Week 24 | -11.84 (20.693) | -10.54 (22.215) | -6.17 (24.224) | -4.00 (19.614)
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 14, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -10.83, 95% CI 2-sided [-12.70 to -8.96], Standard Error of Mean 0.952
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 14, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -7.73, 95% CI 2-sided [-9.58 to -5.87], Standard Error of Mean 0.947
Statistical Analysis 3: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 14, analysis 3]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -9.39, 95% CI 2-sided [-11.33 to -7.45], Standard Error of Mean 0.989
Statistical Analysis 4: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 14, analysis 4]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -7.35, 95% CI 2-sided [-9.29 to -5.42], Standard Error of Mean 0.987
Statistical Analysis 5: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -8.02, 95% CI 2-sided [-9.90 to -6.13], Standard Error of Mean 0.961
Statistical Analysis 6: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -6.46, 95% CI 2-sided [-8.35 to -4.58], Standard Error of Mean 0.960
Statistical Analysis 7: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -7.91, 95% CI 2-sided [-9.88 to -5.93], Standard Error of Mean 1.007
Statistical Analysis 8: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -6.59, 95% CI 2-sided [-8.56 to -4.62], Standard Error of Mean 1.005

27. Secondary Outcome: Change From Baseline in Individual ACR Component: hsCRP at Weeks 36, and 52
Time Frame: Baseline; Weeks 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo to Filgotinib 200 mg | Placebo to Filgotinib 100 mg
Number analyzed (Participants) | 475 | 480 | 325 | 190 | 191
mg/L
  Baseline | 16.13 (21.005) | 16.74 (22.982) | 14.56 (18.003) | 16.54 (24.782) | 15.76 (21.871)
  Change from Baseline at Week 36: number analyzed (Participants) | 408 | 413 | 273 | 179 | 184
  Change from Baseline at Week 36 | -11.51 (21.990) | -10.72 (22.569) | -8.73 (18.214) | -12.12 (23.151) | -8.50 (19.749)
  Change from Baseline at Week 52: number analyzed (Participants) | 396 | 386 | 259 | 169 | 171
  Change from Baseline at Week 52 | -12.19 (20.773) | -11.27 (23.129) | -9.60 (16.511) | -11.43 (20.873) | -8.74 (19.921)

28. Secondary Outcome: Percentage of Participants Who Achieved an Improvement (Decrease) in the HAQ-DI Score ≥ 0.22 at Weeks 2, 4, 12, and 24
Description: The HAQ-DI score is defined as the average of the scores of eight functional categories (dressing and grooming, arising, eating, walking, hygiene, reach, grip, and other activities), usually completed by the participant. Responses in each functional category are collected as 0 (without any difficulty) to 3 (unable to do a task in that area), with or without aids or devices. The eight category scores are averaged into an overall HAQ-DI score on a scale from 0-3 [0 (no disability) to 3 (completely disabled) when 6 or more categories are non-missing, so total possible score is 3. Improvement is defined as reduction in HAQ-DI, (baseline value - postbaseline value) ≥ 0.22. If more than 2 categories are missing, the HAQ-DI score is set to missing. Participants with missing outcomes were set as non-responders.
Time Frame: Weeks 2, 4, 12, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo
Number analyzed (Participants) | 475 | 480 | 325 | 475
percentage of participants
  Week 2: number analyzed (Participants) | 459 | 467 | 316 | 463
  Week 2 | 52.5 [47.8 to 57.2] | 46.7 [42.0 to 51.3] | 51.9 [46.2 to 57.6] | 40.2 [35.6 to 44.7]
  Week 4: number analyzed (Participants) | 459 | 467 | 316 | 463
  Week 4 | 66.2 [61.8 to 70.7] | 58.0 [53.4 to 62.6] | 63.9 [58.5 to 69.4] | 49.9 [45.2 to 54.6]
  Week 12: number analyzed (Participants) | 459 | 467 | 316 | 463
  Week 12 | 78.9 [75.0 to 82.7] | 71.5 [67.3 to 75.7] | 72.8 [67.6 to 77.9] | 57.9 [53.3 to 62.5]
  Week 24: number analyzed (Participants) | 459 | 467 | 316 | 463
  Week 24 | 76.0 [72.0 to 80.0] | 73.4 [69.3 to 77.6] | 71.2 [66.1 to 76.4] | 59.4 [54.8 to 64.0]
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; Filgotinib 200 mg vs Placebo at Week 2; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 12.3, 95% CI 2-sided [5.7 to 18.9]
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; Filgotinib 100 mg vs Placebo at Week 2; Test type: Superiority; p = 0.043, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 6.5, 95% CI 2-sided [-0.1 to 13.1]
Statistical Analysis 3: Comparison: Filgotinib 200 mg vs Placebo; Filgotinib 200 mg vs Placebo at Week 4; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 16.3, 95% CI 2-sided [9.8 to 22.8]
Statistical Analysis 4: Comparison: Filgotinib 100 mg vs Placebo; Filgotinib 100 mg vs Placebo at Week 4; Test type: Superiority; p = 0.011, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 8.1, 95% CI 2-sided [1.5 to 14.7]
Statistical Analysis 5: Comparison: Filgotinib 200 mg vs Placebo; Filgotinib 200 mg vs Placebo at Week 12; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 21.0, 95% CI 2-sided [14.9 to 27.0]
Statistical Analysis 6: Comparison: Filgotinib 100 mg vs Placebo; Filgotinib 100 mg vs Placebo at Week 12; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 13.6, 95% CI 2-sided [7.3 to 19.9]
Statistical Analysis 7: Comparison: Filgotinib 200 mg vs Placebo; Filgotinib 200 mg vs Placebo at Week 24; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 16.6, 95% CI 2-sided [10.5 to 22.8]
Statistical Analysis 8: Comparison: Filgotinib 100 mg vs Placebo; Filgotinib 100 mg vs Placebo at Week 24; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 14.1, 95% CI 2-sided [7.8 to 20.3]

29. Secondary Outcome: Percentage of Participants Who Achieved an Improvement (Decrease) in the HAQ-DI Score ≥ 0.22 at Weeks 36, and 52
Description: as for outcome 28
Time Frame: Weeks 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo to Filgotinib 200 mg | Placebo to Filgotinib 100 mg
Number analyzed (Participants) | 475 | 480 | 325 | 190 | 191
percentage of participants
  Week 36: number analyzed (Participants) | 459 | 467 | 316 | 185 | 188
  Week 36 | 77.1 [73.2 to 81.1] | 74.9 [70.9 to 79.0] | 71.5 [66.4 to 76.7] | 83.2 [77.6 to 88.9] | 77.7 [71.4 to 83.9]
  Week 52: number analyzed (Participants) | 459 | 467 | 316 | 185 | 188
  Week 52 | 75.8 [71.8 to 79.8] | 73.0 [68.9 to 77.2] | 70.3 [65.1 to 75.5] | 81.6 [75.8 to 87.5] | 71.8 [65.1 to 78.5]

30. Secondary Outcome: Change From Baseline in DAS28 (CRP) at Weeks 2, 4, 12, and 24
Description: The DAS28 score is a measure of the participant's disease activity calculated using the tender joint counts (28 joints), swollen joint counts (28 joints), SGA (VAS: 0 = no disease activity to 100 = maximum disease activity), and hsCRP for a total possible score of 1 to 9.4. Higher values indicate higher disease activity. A negative change from baseline indicates improvement.
Time Frame: Baseline; Weeks 2, 4, 12, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo
Number analyzed (Participants) | 475 | 480 | 325 | 475
score on a scale
  Baseline | 5.8 (0.88) | 5.7 (0.95) | 5.7 (0.88) | 5.7 (0.91)
  Change from Baseline at Week 2: number analyzed (Participants) | 452 | 464 | 314 | 461
  Change from Baseline at Week 2 | -1.3 (1.05) | -1.0 (0.90) | -1.1 (0.90) | -0.6 (0.79)
  Change from Baseline at Week 4: number analyzed (Participants) | 463 | 467 | 318 | 454
  Change from Baseline at Week 4 | -1.7 (1.19) | -1.4 (1.07) | -1.4 (1.04) | -0.9 (0.98)
  Change from Baseline at Week 12: number analyzed (Participants) | 455 | 452 | 308 | 431
  Change from Baseline at Week 12 | -2.5 (1.24) | -2.2 (1.17) | -2.2 (1.12) | -1.6 (1.19)
  Change from Baseline at Week 24: number analyzed (Participants) | 415 | 419 | 281 | 368
  Change from Baseline at Week 24 | -3.1 (1.17) | -2.8 (1.08) | -2.7 (1.20) | -2.2 (1.20)
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 14, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.7, 95% CI 2-sided [-0.9 to -0.6], Standard Error of Mean 0.06
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 14, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.4, 95% CI 2-sided [-0.5 to -0.3], Standard Error of Mean 0.06
Statistical Analysis 3: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 14, analysis 3]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.8, 95% CI 2-sided [-0.9 to -0.7], Standard Error of Mean 0.07
Statistical Analysis 4: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 14, analysis 4]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.5, 95% CI 2-sided [-0.7 to -0.4], Standard Error of Mean 0.07
Statistical Analysis 5: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -1.0, 95% CI 2-sided [-1.1 to -0.8], Standard Error of Mean 0.07
Statistical Analysis 6: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.7, 95% CI 2-sided [-0.8 to -0.5], Standard Error of Mean 0.07
Statistical Analysis 7: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -1.0, 95% CI 2-sided [-1.1 to -0.8], Standard Error of Mean 0.08
Statistical Analysis 8: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.7, 95% CI 2-sided [-0.8 to -0.5], Standard Error of Mean 0.08

31. Secondary Outcome: Change From Baseline in DAS28 (CRP) at Weeks 36, and 52
Description: as for outcome 30
Time Frame: Baseline; Weeks 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo to Filgotinib 200 mg | Placebo to Filgotinib 100 mg
Number analyzed (Participants) | 475 | 480 | 325 | 190 | 191
score on a scale
  Baseline | 5.8 (0.88) | 5.7 (0.95) | 5.7 (0.88) | 5.9 (0.89) | 5.6 (0.89)
  Change from Baseline at Week 36: number analyzed (Participants) | 407 | 413 | 272 | 177 | 184
  Change from Baseline at Week 36 | -3.2 (1.09) | -2.9 (1.17) | -2.9 (1.16) | -3.3 (1.10) | -2.8 (1.08)
  Change from Baseline at Week 52: number analyzed (Participants) | 393 | 385 | 259 | 169 | 171
  Change from Baseline at Week 52 | -3.4 (1.11) | -3.1 (1.09) | -3.1 (1.13) | -3.3 (1.16) | -3.0 (1.04)

32. Secondary Outcome: Percentage of Participants Who Achieved DAS28 (CRP) ≤ 3.2 at Weeks 2, 4, and 24
Description: as for outcome 5
Time Frame: Weeks 2, 4, and 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo
Number analyzed (Participants) | 475 | 480 | 325 | 475
percentage of participants
  Week 2 | 13.1 [9.9 to 16.2] | 8.1 [5.6 to 10.7] | 9.8 [6.5 to 13.2] | 3.6 [1.8 to 5.4]
  Week 4 | 25.5 [21.5 to 29.5] | 20.4 [16.7 to 24.1] | 20.9 [16.3 to 25.5] | 9.3 [6.6 to 12.0]
  Week 24 | 60.6 [56.1 to 65.1] | 53.1 [48.6 to 57.7] | 50.5 [44.9 to 56.1] | 33.7 [29.3 to 38.0]
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; Filgotinib 200 mg vs Placebo at Week 2; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 9.5, 95% CI 2-sided [5.8 to 13.1]
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; Filgotinib 100 mg vs Placebo at Week 2; Test type: Superiority; p = 0.004, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 4.5, 95% CI 2-sided [1.4 to 7.7]
Statistical Analysis 3: Comparison: Filgotinib 200 mg vs Placebo; Filgotinib 200 mg vs Placebo at Week 4; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 16.2, 95% CI 2-sided [11.3 to 21.1]
Statistical Analysis 4: Comparison: Filgotinib 100 mg vs Placebo; Filgotinib 100 mg vs Placebo at Week 4; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 11.2, 95% CI 2-sided [6.5 to 15.8]
Statistical Analysis 5: Comparison: Filgotinib 200 mg vs Placebo; Filgotinib 200 mg vs Placebo at Week 24; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 26.9, 95% CI 2-sided [20.6 to 33.3]
Statistical Analysis 6: Comparison: Filgotinib 100 mg vs Placebo; Filgotinib 100 mg vs Placebo at Week 24; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 19.4, 95% CI 2-sided [13.1 to 25.8]

33. Secondary Outcome: Percentage of Participants Who Achieved DAS28 (CRP) ≤ 3.2 at Weeks 36, and 52
Description: as for outcome 5
Time Frame: Weeks 36, and 52
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo to Filgotinib 200 mg | Placebo to Filgotinib 100 mg
Number analyzed (Participants) | 475 | 480 | 325 | 190 | 191
percentage of participants
  Week 36 | 67.4 [63.0 to 71.7] | 60.2 [55.7 to 64.7] | 58.2 [52.6 to 63.7] | 74.7 [68.3 to 81.2] | 66.5 [59.5 to 73.4]
  Week 52 | 68.2 [63.9 to 72.5] | 62.1 [57.6 to 66.5] | 61.8 [56.4 to 67.3] | 69.5 [62.7 to 76.3] | 67.5 [60.6 to 74.4]

34. Secondary Outcome: Percentage of Participants Who Achieved DAS28 (CRP) < 2.6 at Weeks 2, 4, and 24
Description: as for outcome 5
Time Frame: Weeks 2, 4, and 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo
Number analyzed (Participants) | 475 | 480 | 325 | 475
percentage of participants
  Week 2 | 5.1 [3.0 to 7.1] | 1.7 [0.4 to 2.9] | 3.4 [1.3 to 5.5] | 0.6 [0.0 to 1.4]
  Week 4 | 13.7 [10.5 to 16.9] | 8.8 [6.1 to 11.4] | 8.0 [4.9 to 11.1] | 2.9 [1.3 to 4.6]
  Week 24 | 48.4 [43.8 to 53.0] | 35.2 [30.8 to 39.6] | 35.7 [30.3 to 41.1] | 16.2 [12.8 to 19.6]
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; Filgotinib 200 mg vs Placebo at Week 2; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 4.4, 95% CI 2-sided [2.1 to 6.7]
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; Filgotinib 100 mg vs Placebo at Week 2; Test type: Superiority; p = 0.17, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 1.0, 95% CI 2-sided [-0.5 to 2.6]
Statistical Analysis 3: Comparison: Filgotinib 200 mg vs Placebo; Filgotinib 200 mg vs Placebo at Week 4; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 10.7, 95% CI 2-sided [7.1 to 14.4]
Statistical Analysis 4: Comparison: Filgotinib 100 mg vs Placebo; Filgotinib 100 mg vs Placebo at Week 4; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 5.8, 95% CI 2-sided [2.6 to 9.0]
Statistical Analysis 5: Comparison: Filgotinib 200 mg vs Placebo; Filgotinib 200 mg vs Placebo at Week 24; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 32.2, 95% CI 2-sided [26.4 to 38.0]
Statistical Analysis 6: Comparison: Filgotinib 100 mg vs Placebo; Filgotinib 100 mg vs Placebo at Week 24; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 19.0, 95% CI 2-sided [13.4 to 24.6]
Statistical Analysis 7: Comparison: Filgotinib 200 mg vs Adalimumab; Filgotinib 200 mg vs Adalimumab at Week 24; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 12.7, 95% CI 2-sided [5.6 to 19.9]
Statistical Analysis 8: Comparison: Filgotinib 100 mg vs Adalimumab; Filgotinib 100 mg vs Adalimumab at Week 24; Test type: Superiority; p = 0.88, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = -0.5, 95% CI 2-sided [-7.5 to 6.5]
Statistical Analysis 9: Comparison: Filgotinib 200 mg vs Adalimumab; Filgotinib 200 mg vs Adalimumab at Week 24; Test type: Non-Inferiority — For non-inferiority test, the approach proposed by Liu 2014 was used to demonstrate that each filgotinib dose preserves more than 50% of the effect of adalimumab on the response rate of DAS28 (CRP) < 2.6 at using NRI; p < 0.001, Method proposed by [Liu 2014] — P-value of non-inferiority test was calculated from approach proposed by [Liu 2014]
Statistical Analysis 10: Comparison: Filgotinib 100 mg vs Adalimumab; Filgotinib 100 mg vs Adalimumab at Week 24; Test type: Non-Inferiority — [test comment as in outcome 34, analysis 9]; p < 0.001, Method proposed by [Liu 2014] — P-value of non-inferiority test was calculated from approach proposed by [Liu 2014]

35. Secondary Outcome: Percentage of Participants Who Achieved DAS28 (CRP) < 2.6 at Weeks 36, and 52
Description: as for outcome 5
Time Frame: Weeks 36, and 52
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo to Filgotinib 200 mg | Placebo to Filgotinib 100 mg
Number analyzed (Participants) | 475 | 480 | 325 | 190 | 191
percentage of participants
  Week 36 | 50.3 [45.7 to 54.9] | 42.9 [38.4 to 47.4] | 42.5 [36.9 to 48.0] | 52.1 [44.7 to 59.5] | 46.1 [38.7 to 53.4]
  Week 52 | 54.5 [49.9 to 59.1] | 44.8 [40.2 to 49.3] | 48.6 [43.0 to 54.2] | 50.5 [43.2 to 57.9] | 50.8 [43.4 to 58.1]

36. Secondary Outcome: American College of Rheumatology N Percent Improvement (ACR-N) at Weeks 2, 4, 12, and 24
Description: ACR-N is defined as the smallest percentage improvement from baseline in swollen joints, tender joints and the median of the following 5 items (PGA, SGA, subject's pain assessment, HAQ-DI and hsCRP). It has a range between 0 and 100%. PGA and SGA assessed using VAS on a scale of 0-100 [0 and 100 indicating no disease activity and maximum disease activity]; subject's pain assessment using VAS on a scale of 0-100 [0 and 100 indicating no pain and unbearable pain]; HAQ-DI score contains 20 questions,8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities and scored on a scale of 0-3 [0 and 3 indicating without difficulty and unable to do]. If this calculation results in a negative value, then the ACR-N is set to 0. The ACR-N value indicates an improvement of N%, with higher numbers indicating greater improvement.
Time Frame: Weeks 2, 4, 12, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent improvement
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo
Number analyzed (Participants) | 475 | 480 | 325 | 475
percent improvement
  Week 2: number analyzed (Participants) | 441 | 451 | 306 | 450
  Week 2 | 18.3 (19.98) | 14.0 (17.14) | 16.3 (18.41) | 8.0 (12.82)
  Week 4: number analyzed (Participants) | 453 | 453 | 311 | 443
  Week 4 | 27.4 (25.24) | 23.0 (22.26) | 23.8 (22.94) | 15.1 (18.92)
  Week 12: number analyzed (Participants) | 445 | 436 | 300 | 422
  Week 12 | 46.8 (28.46) | 40.6 (27.32) | 40.4 (26.18) | 28.1 (25.22)
  Week 24: number analyzed (Participants) | 402 | 408 | 276 | 360
  Week 24 | 58.8 (27.76) | 55.4 (26.47) | 54.3 (28.13) | 42.6 (27.73)

37. Secondary Outcome: ACR N Percent Improvement (ACR-N) at Weeks 36, and 52
Description: as for outcome 36
Time Frame: Weeks 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent improvement
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo to Filgotinib 200 mg | Placebo to Filgotinib 100 mg
Number analyzed (Participants) | 475 | 480 | 325 | 190 | 191
percent improvement
  Week 36: number analyzed (Participants) | 397 | 406 | 267 | 171 | 181
  Week 36 | 62.5 (26.01) | 59.1 (27.47) | 58.6 (27.17) | 63.2 (24.59) | 56.1 (27.30)
  Week 52: number analyzed (Participants) | 385 | 379 | 255 | 165 | 170
  Week 52 | 66.0 (25.89) | 63.1 (26.34) | 63.5 (27.03) | 63.8 (28.00) | 59.7 (26.81)

38. Secondary Outcome: Number of Participants With European League Against Rheumatism (EULAR) Response at Weeks 2, 4, 12, and 24
Description: Good Response: DAS28(CRP) at visit ≤3.2 and improvement from baseline >1.2. Moderate Response: DAS28(CRP) at visit ≤3.2 and improvement from baseline >0.6 and ≤1.2; DAS28(CRP) at visit >3.2 and ≤5.1 and improvement from baseline >0.6; DAS 28(CRP) at visit >5.1 and improvement from baseline >1.2.
  No Response: DAS28(CRP) at visit ≤5.1 and improvement from baseline ≤0.6; DAS 28(CRP) >5.1 at visit and improvement from baseline ≤1.2.
Time Frame: Weeks 2, 4, 12, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo
Number analyzed (Participants) | 475 | 480 | 325 | 475
Participants
  Week 2: number analyzed (Participants) | 452 | 464 | 314 | 461
  Week 2: Good Response | 58 | 32 | 27 | 15
  Week 2: Moderate Response | 237 | 213 | 158 | 133
  Week 2: No Response | 157 | 219 | 129 | 313
  Week 4: number analyzed (Participants) | 463 | 467 | 318 | 454
  Week 4: Good Response | 117 | 86 | 61 | 37
  Week 4: Moderate Response | 231 | 242 | 156 | 189
  Week 4: No Response | 115 | 139 | 101 | 228
  Week 12: number analyzed (Participants) | 455 | 452 | 308 | 431
  Week 12: Good Response | 234 | 177 | 138 | 106
  Week 12: Moderate Response | 188 | 225 | 138 | 224
  Week 12: No Response | 33 | 50 | 32 | 101
  Week 24: number analyzed (Participants) | 415 | 419 | 281 | 368
  Week 24: Good Response | 284 | 250 | 163 | 154
  Week 24: Moderate Response | 124 | 156 | 97 | 170
  Week 24: No Response | 7 | 13 | 21 | 44

39. Secondary Outcome: Number of Participants With EULAR Response at Weeks 36, and 52
Description: as for outcome 38
Time Frame: Weeks 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo to Filgotinib 200 mg | Placebo to Filgotinib 100 mg
Number analyzed (Participants) | 475 | 480 | 325 | 190 | 191
Participants
  Week 36: number analyzed (Participants) | 407 | 413 | 272 | 177 | 184
  Week 36: Good Response | 306 | 276 | 180 | 139 | 124
  Week 36: Moderate Response | 99 | 126 | 84 | 38 | 54
  Week 36: No Response | 2 | 11 | 8 | 0 | 6
  Week 52: number analyzed (Participants) | 393 | 385 | 259 | 169 | 171
  Week 52: Good Response | 308 | 282 | 189 | 129 | 126
  Week 52: Moderate Response | 82 | 98 | 66 | 38 | 42
  Week 52: No Response | 3 | 5 | 4 | 2 | 3

40. Secondary Outcome: Change From Baseline in Clinical Disease Activity Index (CDAI) at Weeks 2, 4, 12, and 24
Description: CDAI is calculated using formula: CDAI = TJC based on 28 joints (TJC28) + SJC based on 28 joints (SJC28) + SGA + PGA. PGA and SGA are assessed using a VAS on a scale of 0-10 [0 and 10 indicating no disease activity and maximum disease activity]. CDAI can range from 0 to 76, with higher score indicating more severe disease activity status. A negative change from baseline indicates improvement.
Time Frame: Baseline; Weeks 2, 4, 12, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo
Number analyzed (Participants) | 475 | 480 | 325 | 475
score on a scale
  Baseline | 39.5 (11.85) | 38.6 (12.23) | 39.2 (11.51) | 39.6 (11.66)
  Change from Baseline at Week 2: number analyzed (Participants) | 463 | 469 | 315 | 461
  Change from Baseline at Week 2 | -12.7 (11.86) | -10.7 (11.17) | -11.7 (10.06) | -8.2 (10.10)
  Change from Baseline at Week 4: number analyzed (Participants) | 468 | 466 | 317 | 457
  Change from Baseline at Week 4 | -17.6 (12.66) | -15.6 (12.07) | -15.4 (11.13) | -12.4 (11.79)
  Change from Baseline at Week 12: number analyzed (Participants) | 456 | 449 | 308 | 433
  Change from Baseline at Week 12 | -26.0 (12.41) | -23.3 (12.32) | -23.5 (11.43) | -20.3 (13.30)
  Change from Baseline at Week 24: number analyzed (Participants) | 413 | 419 | 283 | 373
  Change from Baseline at Week 24 | -30.6 (11.88) | -28.6 (11.57) | -28.4 (11.45) | -26.3 (12.38)
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 14, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -4.6, 95% CI 2-sided [-5.9 to -3.2], Standard Error of Mean 0.68
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 14, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -3.0, 95% CI 2-sided [-4.3 to -1.6], Standard Error of Mean 0.68
Statistical Analysis 3: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 14, analysis 3]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -5.2, 95% CI 2-sided [-6.6 to -3.8], Standard Error of Mean 0.73
Statistical Analysis 4: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 14, analysis 4]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -3.9, 95% CI 2-sided [-5.3 to -2.4], Standard Error of Mean 0.73
Statistical Analysis 5: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -5.9, 95% CI 2-sided [-7.3 to -4.6], Standard Error of Mean 0.69
Statistical Analysis 6: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -4.4, 95% CI 2-sided [-5.8 to -3.1], Standard Deviation 0.69
Statistical Analysis 7: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -5.7, 95% CI 2-sided [-6.9 to -4.5], Standard Error of Mean 0.62
Statistical Analysis 8: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -4.1, 95% CI 2-sided [-5.3 to -2.9], Standard Error of Mean 0.62

41. Secondary Outcome: Change From Baseline in CDAI at Weeks 36, and 52
Description: CDAI is calculated using formula: CDAI = TJC28 + SJC28 + SGA + PGA. PGA and SGA are assessed using a VAS on a scale of 0-10 [0 and 10 indicating no disease activity and maximum disease activity]. CDAI can range from 0 to 76, with higher score indicating more severe disease activity status. A negative change from baseline indicates improvement.
Time Frame: Baseline; Weeks 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo to Filgotinib 200 mg | Placebo to Filgotinib 100 mg
Number analyzed (Participants) | 475 | 480 | 325 | 190 | 191
score on a scale
  Baseline | 39.5 (11.85) | 38.6 (12.23) | 39.2 (11.51) | 41.4 (11.03) | 37.8 (11.23)
  Change from Baseline at Week 36: number analyzed (Participants) | 409 | 416 | 273 | 176 | 187
  Change from Baseline at Week 36 | -32.1 (11.60) | -29.9 (12.18) | -30.4 (11.21) | -33.8 (11.15) | -29.0 (11.02)
  Change from Baseline at Week 52: number analyzed (Participants) | 399 | 397 | 265 | 173 | 177
  Change from Baseline at Week 52 | -32.9 (11.69) | -30.9 (11.70) | -31.6 (11.44) | -34.0 (11.20) | -30.7 (10.80)

42. Secondary Outcome: Change From Baseline in Simplified Disease Activity Index (SDAI) at Weeks 2, 4, 12, and 24
Description: SDAI is a composite measure that sums the TJC28, SJC28, SGA, PGA, and the hsCRP (in mg/dL). PGA and SGA assessed using VAS on a scale of 0-10 [0 and 10 indicating no disease activity and maximum disease activity]. Higher score indicates more severe disease activity status and total possible score is 0 to 86. A negative change from baseline indicates improvement.
Time Frame: Baseline; Weeks 2, 4, 12, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo
Number analyzed (Participants) | 475 | 480 | 325 | 475
score on a scale
  Baseline | 41.2 (12.26) | 40.2 (12.79) | 40.6 (11.88) | 41.2 (12.37)
  Change from Baseline at Week 2: number analyzed (Participants) | 451 | 460 | 312 | 458
  Change from Baseline at Week 2 | -14.0 (12.19) | -11.4 (11.41) | -12.5 (10.52) | -8.2 (10.38)
  Change from Baseline at Week 4: number analyzed (Participants) | 462 | 462 | 316 | 450
  Change from Baseline at Week 4 | -18.6 (13.08) | -16.4 (12.31) | -16.1 (11.47) | -12.5 (12.18)
  Change from Baseline at Week 12: number analyzed (Participants) | 454 | 444 | 305 | 429
  Change from Baseline at Week 12 | -27.1 (12.69) | -24.1 (12.54) | -24.3 (12.03) | -20.6 (13.85)
  Change from Baseline at Week 24: number analyzed (Participants) | 410 | 415 | 281 | 366
  Change from Baseline at Week 24 | -31.8 (12.18) | -29.7 (12.01) | -29.0 (12.19) | -26.6 (12.91)
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 14, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -5.7, 95% CI 2-sided [-7.1 to -4.4], Standard Error of Mean 0.70
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 14, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -3.6, 95% CI 2-sided [-5.0 to -2.2], Standard Error of Mean 0.70
Statistical Analysis 3: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 14, analysis 3]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -6.1, 95% CI 2-sided [-7.6 to -4.6], Standard Error of Mean 0.75
Statistical Analysis 4: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 14, analysis 4]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -4.5, 95% CI 2-sided [-6.0 to -3.1], Standard Error of Mean 0.75
Statistical Analysis 5: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -6.8, 95% CI 2-sided [-8.2 to -5.4], Standard Error of Mean 0.71
Statistical Analysis 6: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -5.1, 95% CI 2-sided [-6.5 to -3.7], Standard Error of Mean 0.71
Statistical Analysis 7: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -6.5, 95% CI 2-sided [-7.8 to -5.3], Standard Error of Mean 0.65
Statistical Analysis 8: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -4.8, 95% CI 2-sided [-6.1 to -3.5], Standard Error of Mean 0.65

43. Secondary Outcome: Change From Baseline in SDAI at Weeks 36, and 52
Description: as for outcome 42
Time Frame: Baseline; Weeks 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo to Filgotinib 200 mg | Placebo to Filgotinib 100 mg
Number analyzed (Participants) | 475 | 480 | 325 | 190 | 191
score on a scale
  Baseline | 41.2 (12.26) | 40.2 (12.79) | 40.6 (11.88) | 43.0 (11.81) | 39.4 (11.81)
  Change from Baseline at Week 36: number analyzed (Participants) | 405 | 412 | 271 | 175 | 183
  Change from Baseline at Week 36 | -33.3 (11.92) | -31.0 (12.69) | -31.2 (11.73) | -35.1 (11.83) | -29.9 (11.40)
  Change from Baseline at Week 52: number analyzed (Participants) | 393 | 385 | 259 | 169 | 171
  Change from Baseline at Week 52 | -34.1 (12.15) | -32.0 (12.25) | -32.6 (11.99) | -34.9 (11.83) | -31.6 (11.11)

44. Secondary Outcome: Change From Baseline in mTSS at Week 52
Description: as for outcome 4
Time Frame: Baseline; Week 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo to Filgotinib 200 mg | Placebo to Filgotinib 100 mg
Number analyzed (Participants) | 468 | 472 | 319 | 187 | 188
score on a scale
  Baseline | 32.62 (48.306) | 36.24 (52.956) | 33.94 (53.803) | 26.68 (45.870) | 32.38 (55.012)
  Change from Baseline at Week 52: number analyzed (Participants) | 417 | 411 | 273 | 180 | 178
  Change from Baseline at Week 52 | 0.21 (1.434) | 0.50 (2.098) | 0.58 (3.621) | 0.63 (2.782) | 0.90 (3.152)
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo to Filgotinib 200 mg; LS-Mean, 95% CI, and P-value were provided from MMRM. Missing change scores were not imputed using the MMRM approach assuming an unstructured variance-covariance matrix for the repeated measures; Test type: Superiority; p = 0.042, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.39, 95% CI 2-sided [-0.77 to -0.01]
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo to Filgotinib 100 mg; [analysis description as in outcome 44, analysis 1]; Test type: Superiority; p = 0.039, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.39, 95% CI 2-sided [-0.77 to -0.02]

45. Secondary Outcome: Percentage of Participants With no Radiographic Progression From Baseline at Week 24
Description: Participant's radiographs of bilateral hands, wrists and feet are taken and evaluated through central review using the mTSS method. No radiographic progression is defined by the change from baseline in mTSS and is reported for the following categories: Change in mTSS ≤ 0.5, Change in mTSS ≤ 0 and Change in mTSS ≤ smallest detectable change (SDC).
Time Frame: Baseline; Weeks 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo
Number analyzed (Participants) | 475 | 480 | 325 | 475
percentage of participants
  Change in mTSS ≤ 0.5: number analyzed (Participants) | 405 | 404 | 271 | 351
  Change in mTSS ≤ 0.5 | 93.8 [91.4 to 96.3] | 91.1 [88.2 to 94.0] | 91.9 [88.4 to 95.3] | 87.2 [83.5 to 90.8]
  Change in mTSS ≤ 0: number analyzed (Participants) | 405 | 404 | 271 | 351
  Change in mTSS ≤ 0 | 87.9 [84.6 to 91.2] | 85.9 [82.4 to 89.4] | 86.3 [82.1 to 90.6] | 80.9 [76.7 to 85.2]
  Change in mTSS ≤ SDC (1.36): number analyzed (Participants) | 405 | 404 | 271 | 351
  Change in mTSS ≤ SDC (1.36) | 95.8 [93.7 to 97.9] | 95.0 [92.8 to 97.3] | 94.5 [91.6 to 97.4] | 90.3 [87.1 to 93.6]
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; Filgotinib 200 mg vs Placebo at Week 24 for change in mTSS ≤ 0.5; Test type: Superiority; p = 0.002, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in non-progression rate = 6.6, 95% CI 2-sided [2.2 to 11.1]
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; Filgotinib 100 mg vs Placebo at Week 24 for change in mTSS ≤ 0.5; Test type: Superiority; p = 0.073, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in non-progression rate = 3.9, 95% CI 2-sided [-0.8 to 8.6]
Statistical Analysis 3: Comparison: Filgotinib 200 mg vs Placebo; Filgotinib 200 mg vs Placebo at Week 24 for change in mTSS ≤ 0; Test type: Superiority; p = 0.009, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in non-progression rate = 7.0, 95% CI 2-sided [1.5 to 12.5]
Statistical Analysis 4: Comparison: Filgotinib 100 mg vs Placebo; Filgotinib 100 mg vs Placebo at Week 24 for change in mTSS ≤ 0; Test type: Superiority; p = 0.061, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in non-progression rate = 5.0, 95% CI 2-sided [-0.6 to 10.6]
Statistical Analysis 5: Comparison: Filgotinib 200 mg vs Placebo; Filgotinib 200 mg vs Placebo at Week 24 for change in mTSS ≤ SDC (1.36); Test type: Superiority; p = 0.004, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in non-progression rate = 5.5, 95% CI 2-sided [1.6 to 9.4]
Statistical Analysis 6: Comparison: Filgotinib 100 mg vs Placebo; Filgotinib 100 mg vs Placebo at Week 24 for change in mTSS ≤ SDC (1.36); Test type: Superiority; p = 0.012, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in non-progression rate = 4.7, 95% CI 2-sided [0.7 to 8.8]

46. Secondary Outcome: Percentage of Participants With no Radiographic Progression From Baseline at Week 52
Description: as for outcome 45
Time Frame: Baseline; Week 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo to Filgotinib 200 mg | Placebo to Filgotinib 100 mg
Number analyzed (Participants) | 475 | 480 | 325 | 190 | 191
percentage of participants
  Change in mTSS ≤ 0.5: number analyzed (Participants) | 417 | 411 | 273 | 180 | 178
  Change in mTSS ≤ 0.5 | 92.1 [89.4 to 94.8] | 87.1 [83.7 to 90.5] | 88.6 [84.7 to 92.6] | 83.9 [78.2 to 89.5] | 83.7 [78.0 to 89.4]
  Change in mTSS ≤ 0: number analyzed (Participants) | 417 | 411 | 273 | 180 | 178
  Change in mTSS ≤ 0 | 87.5 [84.2 to 90.8] | 81.3 [77.4 to 85.2] | 82.4 [77.7 to 87.1] | 73.3 [66.6 to 80.1] | 77.0 [70.5 to 83.4]
  Change in mTSS ≤ SDC (1.83): number analyzed (Participants) | 417 | 411 | 273 | 180 | 178
  Change in mTSS ≤ SDC (1.83) | 95.0 [92.7 to 97.2] | 91.5 [88.7 to 94.3] | 94.1 [91.2 to 97.1] | 90.0 [85.3 to 94.7] | 87.6 [82.5 to 92.8]

47. Secondary Outcome: 36-Item Short Form Survey (SF-36) Physical Component Summary (PCS) Score at Weeks 4, 12, and 24
Description: The SF-36 is a 36-item, self-reported, generic, comprehensive, and health-related quality of life questionnaire based on 8 health domains in 2 components: physical well-being (physical functioning, role-physical, bodily pain, general health perceptions), mental well-being (vitality, social functioning, role-emotional, and mental health). Each domain is scored by summing the individual items and transforming the scores into a 0 to 100 scale with highest possible score of 100. Higher scores indicate better health status or functioning.
Time Frame: Weeks 4, 12, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo
Number analyzed (Participants) | 475 | 480 | 325 | 475
score on a scale
  Week 4: number analyzed (Participants) | 471 | 475 | 321 | 465
  Week 4 | 39.0 (8.22) | 38.2 (8.35) | 37.7 (8.07) | 36.1 (7.40)
  Week 12: number analyzed (Participants) | 461 | 464 | 312 | 441
  Week 12 | 42.7 (8.30) | 42.1 (8.69) | 41.3 (8.57) | 38.8 (7.83)
  Week 24: number analyzed (Participants) | 426 | 427 | 285 | 376
  Week 24 | 43.9 (8.49) | 43.7 (8.64) | 43.2 (8.95) | 40.7 (8.10)

48. Secondary Outcome: SF-36 PCS Score at Weeks 36, and 52
Description: as for outcome 47
Time Frame: Weeks 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo to Filgotinib 200 mg | Placebo to Filgotinib 100 mg
Number analyzed (Participants) | 475 | 480 | 325 | 190 | 191
score on a scale
  Week 36: number analyzed (Participants) | 413 | 417 | 276 | 181 | 188
  Week 36 | 45.2 (8.28) | 44.4 (8.54) | 43.8 (8.84) | 45.2 (7.99) | 43.2 (8.82)
  Week 52: number analyzed (Participants) | 400 | 399 | 267 | 174 | 180
  Week 52 | 45.6 (8.35) | 45.1 (8.57) | 45.2 (8.55) | 45.1 (8.26) | 44.1 (8.88)

49. Secondary Outcome: Change From Baseline in SF-36 PCS Score at Weeks 4, and 24
Description: as for outcome 6
Time Frame: Baseline; Weeks 4, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo
Number analyzed (Participants) | 473 | 479 | 323 | 474
score on a scale
  Baseline | 33.4 (7.17) | 33.6 (7.75) | 32.8 (7.74) | 32.9 (7.11)
  Change from Baseline at Week 4: number analyzed (Participants) | 469 | 474 | 319 | 464
  Change from Baseline at Week 4 | 5.6 (6.57) | 4.6 (6.50) | 5.0 (6.65) | 3.1 (6.32)
  Change from Baseline at Week 24: number analyzed (Participants) | 424 | 426 | 283 | 376
  Change from Baseline at Week 24 | 10.4 (8.49) | 10.3 (8.64) | 10.4 (8.47) | 7.7 (7.97)
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 14, analysis 3]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 2.7, 95% CI 2-sided [1.9 to 3.4], Standard Error of Mean 0.40
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 14, analysis 4]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 1.7, 95% CI 2-sided [1.0 to 2.5], Standard Error of Mean 0.40
Statistical Analysis 3: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 3.1, 95% CI 2-sided [2.1 to 4.1], Standard Error of Mean 0.52
Statistical Analysis 4: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 3.1, 95% CI 2-sided [2.0 to 4.1], Standard Error of Mean 0.52

50. Secondary Outcome: Change From Baseline in SF-36 PCS Score at Weeks 36, and 52
Description: as for outcome 6
Time Frame: Baseline; Weeks 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo to Filgotinib 200 mg | Placebo to Filgotinib 100 mg
Number analyzed (Participants) | 473 | 479 | 323 | 190 | 191
score on a scale
  Baseline | 33.4 (7.17) | 33.6 (7.75) | 32.8 (7.74) | 32.2 (6.96) | 33.7 (6.96)
  Change from Baseline at Week 36: number analyzed (Participants) | 412 | 416 | 274 | 181 | 188
  Change from Baseline at Week 36 | 11.6 (8.28) | 11.0 (8.53) | 11.1 (9.07) | 12.9 (8.92) | 9.5 (8.13)
  Change from Baseline at Week 52: number analyzed (Participants) | 399 | 398 | 265 | 174 | 180
  Change from Baseline at Week 52 | 12.0 (8.73) | 11.5 (8.74) | 12.4 (9.21) | 13.0 (9.58) | 10.4 (8.05)

51. Secondary Outcome: SF-36 Mental Component Summary (MCS) Score at Weeks 4, 12, and 24
Description: as for outcome 47
Time Frame: Weeks 4, 12, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo
Number analyzed (Participants) | 475 | 480 | 325 | 475
score on a scale
  Week 4: number analyzed (Participants) | 471 | 475 | 321 | 465
  Week 4 | 47.8 (9.90) | 47.9 (9.63) | 47.9 (10.04) | 45.8 (10.35)
  Week 12: number analyzed (Participants) | 460 | 464 | 312 | 441
  Week 12 | 49.3 (9.14) | 49.9 (8.90) | 48.9 (10.28) | 47.7 (10.16)
  Week 24: number analyzed (Participants) | 426 | 427 | 285 | 376
  Week 24 | 50.0 (8.82) | 50.2 (8.93) | 49.3 (10.26) | 49.2 (9.90)

52. Secondary Outcome: SF-36 MCS Score at Weeks 36, and 52
Description: as for outcome 47
Time Frame: Weeks 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo to Filgotinib 200 mg | Placebo to Filgotinib 100 mg
Number analyzed (Participants) | 475 | 480 | 325 | 190 | 191
score on a scale
  Week 36: number analyzed (Participants) | 413 | 417 | 276 | 181 | 188
  Week 36 | 50.1 (8.96) | 51.3 (8.88) | 50.7 (9.67) | 50.7 (9.04) | 50.3 (9.47)
  Week 52: number analyzed (Participants) | 400 | 399 | 267 | 174 | 180
  Week 52 | 50.6 (9.30) | 51.5 (8.99) | 50.8 (9.51) | 50.8 (8.55) | 50.1 (9.21)

53. Secondary Outcome: Change From Baseline in SF-36 MCS Score at Weeks 4, 12, and 24
Description: as for outcome 6
Time Frame: Baseline; Weeks 4, 12, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo
Number analyzed (Participants) | 473 | 479 | 323 | 474
score on a scale
  Baseline | 43.9 (10.44) | 44.6 (10.44) | 44.1 (10.44) | 43.4 (11.01)
  Change from Baseline at Week 4: number analyzed (Participants) | 469 | 474 | 319 | 464
  Change from Baseline at Week 4 | 3.9 (7.96) | 3.4 (8.35) | 3.7 (7.66) | 2.3 (8.72)
  Change from Baseline at Week 12: number analyzed (Participants) | 458 | 463 | 310 | 440
  Change from Baseline at Week 12 | 5.4 (9.45) | 5.4 (8.97) | 4.9 (9.69) | 4.1 (9.50)
  Change from Baseline at Week 24: number analyzed (Participants) | 424 | 426 | 283 | 376
  Change from Baseline at Week 24 | 6.1 (9.23) | 5.7 (9.57) | 5.3 (9.25) | 5.6 (10.28)
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 14, analysis 3]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 1.8, 95% CI 2-sided [0.9 to 2.8], Standard Error of Mean 0.48
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 14, analysis 4]; Test type: Superiority; p = 0.002, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 1.5, 95% CI 2-sided [0.6 to 2.5], Standard Error of Mean 0.48
Statistical Analysis 3: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.006, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 1.5, 95% CI 2-sided [0.4 to 2.5], Standard Error of Mean 0.52
Statistical Analysis 4: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 1.7, 95% CI 2-sided [0.7 to 2.7], Standard Error of Mean 0.52
Statistical Analysis 5: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.086, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 0.9, 95% CI 2-sided [-0.1 to 2.0], Standard Error of Mean 0.55
Statistical Analysis 6: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p = 0.12, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 0.9, 95% CI 2-sided [-0.2 to 1.9], Standard Error of Mean 0.55

54. Secondary Outcome: Change From Baseline in SF-36 MCS Score at Weeks 36, and 52
Description: as for outcome 6
Time Frame: Baseline; Weeks 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo to Filgotinib 200 mg | Placebo to Filgotinib 100 mg
Number analyzed (Participants) | 473 | 479 | 323 | 190 | 191
score on a scale
  Baseline | 43.9 (10.44) | 44.6 (10.44) | 44.1 (10.44) | 43.9 (11.06) | 43.4 (11.03)
  Change from Baseline at Week 36: number analyzed (Participants) | 412 | 416 | 274 | 181 | 188
  Change from Baseline at Week 36 | 6.2 (10.03) | 6.6 (10.46) | 6.6 (9.40) | 6.9 (12.05) | 6.8 (9.84)
  Change from Baseline at Week 52: number analyzed (Participants) | 399 | 398 | 265 | 174 | 180
  Change from Baseline at Week 52 | 6.7 (10.53) | 6.9 (10.61) | 6.7 (9.90) | 7.2 (11.31) | 6.5 (10.35)

55. Secondary Outcome: Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Score at Weeks 4, 12, and 24
Description: FACIT-Fatigue scale is a brief, 13-item, symptom-specific questionnaire that specifically assesses the self-reported severity of fatigue and its impact upon daily activities and functioning in the past 7 days. The FACIT-Fatigue uses 0 (not at all) to 4 (very much) numeric rating scales for a total possible score of 0 to 52.
Time Frame: Weeks 4, 12, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo
Number analyzed (Participants) | 475 | 480 | 325 | 475
score on a scale
  Week 4: number analyzed (Participants) | 468 | 471 | 319 | 457
  Week 4 | 33.9 (10.32) | 33.3 (9.76) | 32.9 (10.11) | 30.9 (10.43)
  Week 12: number analyzed (Participants) | 455 | 457 | 307 | 437
  Week 12 | 36.8 (9.64) | 36.7 (9.67) | 36.1 (9.68) | 33.9 (10.32)
  Week 24: number analyzed (Participants) | 416 | 419 | 277 | 372
  Week 24 | 38.5 (9.17) | 38.5 (8.74) | 37.6 (9.82) | 35.8 (9.94)

56. Secondary Outcome: FACIT-Fatigue Score at Weeks 36, and 52
Description: as for outcome 55
Time Frame: Weeks 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo to Filgotinib 200 mg | Placebo to Filgotinib 100 mg
Number analyzed (Participants) | 475 | 480 | 325 | 190 | 191
score on a scale
  Week 36: number analyzed (Participants) | 395 | 405 | 270 | 177 | 184
  Week 36 | 38.9 (8.84) | 39.5 (8.73) | 38.6 (9.45) | 39.6 (8.78) | 37.4 (9.88)
  Week 52: number analyzed (Participants) | 386 | 379 | 257 | 167 | 174
  Week 52 | 39.8 (8.64) | 39.8 (8.54) | 38.9 (9.87) | 39.4 (8.78) | 38.0 (9.77)

57. Secondary Outcome: Change From Baseline in FACIT-Fatigue Score at Weeks 4, and 24
Description: as for outcome 7
Time Frame: Baseline; Weeks 4, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo
Number analyzed (Participants) | 472 | 477 | 319 | 469
score on a scale
  Baseline | 27.6 (10.68) | 27.8 (10.60) | 27.2 (10.20) | 26.9 (10.34)
  Change from Baseline at Week 4: number analyzed (Participants) | 465 | 470 | 316 | 455
  Change from Baseline at Week 4 | 6.3 (8.59) | 5.7 (8.77) | 5.7 (8.47) | 3.8 (8.76)
  Change from Baseline at Week 24: number analyzed (Participants) | 413 | 417 | 273 | 369
  Change from Baseline at Week 24 | 10.5 (10.63) | 10.8 (10.77) | 10.3 (9.67) | 8.4 (10.48)
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 14, analysis 3]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 2.8, 95% CI 2-sided [1.8 to 3.8], Standard Error of Mean 0.51
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 14, analysis 4]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 2.2, 95% CI 2-sided [1.2 to 3.2], Standard Error of Mean 0.51
Statistical Analysis 3: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 2.6, 95% CI 2-sided [1.5 to 3.8], Standard Error of Mean 0.59
Statistical Analysis 4: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 2.8, 95% CI 2-sided [1.6 to 3.9], Standard Error of Mean 0.59

58. Secondary Outcome: Change From Baseline in FACIT-Fatigue Score at Weeks 36, and 52
Description: as for outcome 7
Time Frame: Baseline; Weeks 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo to Filgotinib 200 mg | Placebo to Filgotinib 100 mg
Number analyzed (Participants) | 472 | 477 | 319 | 189 | 189
score on a scale
  Baseline | 27.6 (10.68) | 27.8 (10.60) | 27.2 (10.20) | 26.8 (10.13) | 27.9 (10.56)
  Change from Baseline at Week 36: number analyzed (Participants) | 393 | 403 | 268 | 176 | 182
  Change from Baseline at Week 36 | 11.0 (10.22) | 11.7 (10.90) | 11.3 (10.18) | 12.8 (10.76) | 9.5 (10.25)
  Change from Baseline at Week 52: number analyzed (Participants) | 384 | 376 | 254 | 166 | 172
  Change from Baseline at Week 52 | 11.9 (10.21) | 12.2 (10.88) | 11.7 (10.79) | 12.9 (11.55) | 10.1 (10.06)

59. Secondary Outcome: Number of Participants by European Quality of Life 5 Dimensions (EQ-5D) Health Profile Categories at Weeks 4, 12, and 24
Description: The EQ-5D-5 levels (EQ-5D-5L) is a standardized measure of health status of the participant at the visit (same day) that provides a simple, generic measure of health for clinical and economic appraisal. EQ-5D-5L consists of 2 components: a descriptive system of the participant's health and a rating of his or her current health state on a 0-100 VAS. The descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. Rating gets recorded on a vertical VAS in which the endpoints are labeled best imaginable health state is 100 (on the top) and worst imaginable health state is 0 (on the bottom). Higher scores of EQ VAS indicate better health.
Time Frame: Weeks 4, 12, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo
Number analyzed (Participants) | 475 | 480 | 325 | 475
Participants
  Mobility: Week 4: number analyzed (Participants) | 468 | 471 | 319 | 457
  Mobility: Week 4: No Problems | 130 | 129 | 84 | 100
  Mobility: Week 4: Slight Problems | 176 | 173 | 107 | 149
  Mobility: Week 4: Moderate Problems | 113 | 122 | 96 | 150
  Mobility: Week 4: Severe Problems | 44 | 46 | 31 | 56
  Mobility: Week 4: Extreme Problems | 5 | 1 | 1 | 2
  Mobility: Week 12: number analyzed (Participants) | 455 | 457 | 307 | 437
  Mobility: Week 12: No Problems | 178 | 177 | 116 | 132
  Mobility: Week 12: Slight Problems | 153 | 151 | 103 | 154
  Mobility: Week 12: Moderate Problems | 99 | 97 | 67 | 112
  Mobility: Week 12: Severe Problems | 21 | 31 | 21 | 38
  Mobility: Week 12: Extreme Problems | 4 | 1 | 0 | 1
  Mobility: week 24: number analyzed (Participants) | 416 | 419 | 277 | 372
  Mobility: week 24: No Problems | 182 | 189 | 117 | 131
  Mobility: week 24: Slight Problems | 142 | 136 | 90 | 126
  Mobility: week 24: Moderate Problems | 68 | 75 | 57 | 89
  Mobility: week 24: Severe Problems | 19 | 17 | 12 | 24
  Mobility: week 24: Extreme Problems | 5 | 2 | 1 | 2
  Self-care: Week 4: number analyzed (Participants) | 468 | 471 | 319 | 457
  Self-care: Week 4: No Problems | 177 | 163 | 111 | 138
  Self-care: Week 4: Slight Problems | 180 | 183 | 120 | 164
  Self-care: Week 4: Moderate Problems | 86 | 103 | 74 | 124
  Self-care: Week 4: Severe Problems | 23 | 20 | 13 | 25
  Self-care: Week 4: Extreme Problems | 2 | 2 | 1 | 6
  Self-care: Week 12: number analyzed (Participants) | 455 | 457 | 307 | 437
  Self-care: Week 12: No Problems | 243 | 222 | 147 | 165
  Self-care: Week 12: Slight Problems | 149 | 150 | 102 | 159
  Self-care: Week 12: Moderate Problems | 53 | 74 | 49 | 88
  Self-care: Week 12: Severe Problems | 8 | 9 | 9 | 21
  Self-care: Week 12: Extreme Problems | 2 | 2 | 0 | 4
  Self-care: Week 24: number analyzed (Participants) | 416 | 419 | 277 | 372
  Self-care: Week 24: No Problems | 255 | 249 | 157 | 164
  Self-care: Week 24: Slight Problems | 109 | 121 | 75 | 140
  Self-care: Week 24: Moderate Problems | 45 | 39 | 36 | 54
  Self-care: Week 24: Severe Problems | 4 | 8 | 7 | 14
  Self-care: Week 24: Extreme Problems | 3 | 2 | 2 | 0
  Usual Activities: Week 4: number analyzed (Participants) | 468 | 471 | 319 | 457
  Usual Activities: Week 4: No Problems | 110 | 102 | 69 | 65
  Usual Activities: Week 4: Slight Problems | 203 | 193 | 133 | 195
  Usual Activities: Week 4: Moderate Problems | 111 | 142 | 90 | 143
  Usual Activities: Week 4: Severe Problems | 38 | 33 | 25 | 52
  Usual Activities: Week 4: Extreme Problems | 6 | 1 | 2 | 2
  Usual Activities: Week 12: number analyzed (Participants) | 455 | 457 | 307 | 437
  Usual Activities: Week 12: No Problems | 157 | 149 | 97 | 103
  Usual Activities: Week 12: Slight Problems | 200 | 191 | 130 | 184
  Usual Activities: Week 12: Moderate Problems | 80 | 90 | 67 | 116
  Usual Activities: Week 12: Severe Problems | 16 | 23 | 13 | 32
  Usual Activities: Week 12: Extreme Problems | 2 | 4 | 0 | 2
  Usual Activities: Week 24: number analyzed (Participants) | 416 | 419 | 277 | 372
  Usual Activities: Week 24: No Problems | 184 | 175 | 109 | 107
  Usual Activities: Week 24: Slight Problems | 164 | 171 | 105 | 163
  Usual Activities: Week 24: Moderate Problems | 54 | 63 | 52 | 86
  Usual Activities: Week 24: Severe Problems | 13 | 9 | 9 | 15
  Usual Activities: Week 24: Extreme Problems | 1 | 1 | 2 | 1
  Pain/Discomfort: Week 4: number analyzed (Participants) | 468 | 471 | 319 | 457
  Pain/Discomfort: Week 4: No Problems | 42 | 38 | 26 | 14
  Pain/Discomfort: Week 4: Slight Problems | 215 | 185 | 118 | 157
  Pain/Discomfort: Week 4: Moderate Problems | 154 | 204 | 127 | 198
  Pain/Discomfort: Week 4: Severe Problems | 51 | 41 | 47 | 80
  Pain/Discomfort: Week 4: Extreme Problems | 6 | 3 | 1 | 8
  Pain/Discomfort: Week 12: number analyzed (Participants) | 455 | 457 | 307 | 437
  Pain/Discomfort: Week 12: No Problems | 58 | 71 | 34 | 29
  Pain/Discomfort: Week 12: Slight Problems | 260 | 217 | 145 | 200
  Pain/Discomfort: Week 12: Moderate Problems | 117 | 150 | 106 | 154
  Pain/Discomfort: Week 12: Severe Problems | 20 | 17 | 22 | 51
  Pain/Discomfort: Week 12: Extreme Problems | 0 | 2 | 0 | 3
  Pain/Discomfort: Week 24: number analyzed (Participants) | 416 | 419 | 277 | 372
  Pain/Discomfort: Week 24: No Problems | 82 | 78 | 56 | 39
  Pain/Discomfort: Week 24: Slight Problems | 226 | 224 | 127 | 196
  Pain/Discomfort: Week 24: Moderate Problems | 86 | 103 | 82 | 110
  Pain/Discomfort: Week 24: Severe Problems | 21 | 13 | 12 | 27
  Pain/Discomfort: Week 24: Extreme Problems | 1 | 1 | 0 | 0
  Anxiety/Depression: Week 4: number analyzed (Participants) | 468 | 471 | 319 | 457
  Anxiety/Depression: Week 4: No Problems | 211 | 224 | 151 | 196
  Anxiety/Depression: Week 4: Slight Problems | 163 | 158 | 111 | 149
  Anxiety/Depression: Week 4: Moderate Problems | 72 | 81 | 44 | 86
  Anxiety/Depression: Week 4: Severe Problems | 21 | 8 | 13 | 25
  Anxiety/Depression: Week 4: Extreme Problems | 1 | 0 | 0 | 1
  Anxiety/Depression: Week 12: number analyzed (Participants) | 455 | 457 | 307 | 437
  Anxiety/Depression: Week 12: No Problems | 235 | 246 | 152 | 216
  Anxiety/Depression: Week 12: Slight Problems | 154 | 143 | 106 | 137
  Anxiety/Depression: Week 12: Moderate Problems | 54 | 63 | 44 | 62
  Anxiety/Depression: Week 12: Severe Problems | 12 | 5 | 4 | 19
  Anxiety/Depression: Week 12: Extreme Problems | 0 | 0 | 1 | 3
  Anxiety/Depression: Week 24: number analyzed (Participants) | 416 | 419 | 277 | 372
  Anxiety/Depression: Week 24: No Problems | 230 | 256 | 160 | 204
  Anxiety/Depression: Week 24: Slight Problems | 136 | 119 | 75 | 120
  Anxiety/Depression: Week 24: Moderate Problems | 42 | 37 | 33 | 39
  Anxiety/Depression: Week 24: Severe Problems | 8 | 5 | 6 | 8
  Anxiety/Depression: Week 24: Extreme Problems | 0 | 2 | 3 | 1

60. Secondary Outcome: Number of Participants by EQ-5D Health Profile Categories at Weeks 36, and 52
Description: as for outcome 59
Time Frame: Weeks 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo to Filgotinib 200 mg | Placebo to Filgotinib 100 mg
Number analyzed (Participants) | 475 | 480 | 325 | 190 | 191
Participants
  Mobility: Week 36: number analyzed (Participants) | 395 | 405 | 270 | 177 | 184
  Mobility: Week 36: No Problems | 202 | 189 | 122 | 86 | 78
  Mobility: Week 36: Slight Problems | 121 | 136 | 82 | 58 | 67
  Mobility: Week 36: Moderate Problems | 58 | 64 | 48 | 26 | 28
  Mobility: Week 36: Severe Problems | 13 | 15 | 16 | 7 | 11
  Mobility: Week 36: Extreme Problems | 1 | 1 | 2 | 0 | 0
  Mobility: Week 52: number analyzed (Participants) | 386 | 379 | 257 | 167 | 174
  Mobility: Week 52: No Problems | 197 | 187 | 130 | 82 | 77
  Mobility: Week 52: Slight Problems | 117 | 115 | 79 | 47 | 61
  Mobility: Week 52: Moderate Problems | 57 | 58 | 38 | 34 | 27
  Mobility: Week 52: Severe Problems | 11 | 19 | 10 | 3 | 8
  Mobility: Week 52: Extreme Problems | 4 | 0 | 0 | 1 | 1
  Self-care: Week 36: number analyzed (Participants) | 395 | 405 | 270 | 177 | 184
  Self-care: Week 36: No Problems | 254 | 249 | 164 | 114 | 108
  Self-care: Week 36: Slight Problems | 104 | 113 | 67 | 45 | 46
  Self-care: Week 36: Moderate Problems | 31 | 36 | 30 | 17 | 25
  Self-care: Week 36: Severe Problems | 5 | 5 | 6 | 1 | 5
  Self-care: Week 36: Extreme Problems | 1 | 2 | 3 | 0 | 0
  Self-care: Week 52: number analyzed (Participants) | 386 | 379 | 257 | 167 | 174
  Self-care: Week 52: No Problems | 251 | 245 | 159 | 105 | 101
  Self-care: Week 52: Slight Problems | 98 | 102 | 72 | 44 | 48
  Self-care: Week 52: Moderate Problems | 30 | 25 | 24 | 16 | 18
  Self-care: Week 52: Severe Problems | 5 | 6 | 2 | 1 | 6
  Self-care: Week 52: Extreme Problems | 2 | 1 | 0 | 1 | 1
  Usual Activities: Week 36: number analyzed (Participants) | 395 | 405 | 270 | 177 | 184
  Usual Activities: Week 36: No Problems | 176 | 172 | 125 | 82 | 72
  Usual Activities: Week 36: Slight Problems | 160 | 171 | 90 | 71 | 70
  Usual Activities: Week 36: Moderate Problems | 50 | 52 | 46 | 21 | 36
  Usual Activities: Week 36: Severe Problems | 7 | 9 | 7 | 3 | 5
  Usual Activities: Week 36: Extreme Problems | 2 | 1 | 2 | 0 | 1
  Usual Activities: Week 52: number analyzed (Participants) | 386 | 379 | 257 | 167 | 174
  Usual Activities: Week 52: No Problems | 183 | 177 | 121 | 75 | 71
  Usual Activities: Week 52: Slight Problems | 151 | 147 | 87 | 64 | 72
  Usual Activities: Week 52: Moderate Problems | 40 | 41 | 42 | 22 | 19
  Usual Activities: Week 52: Severe Problems | 8 | 12 | 6 | 5 | 12
  Usual Activities: Week 52: Extreme Problems | 4 | 2 | 1 | 1 | 0
  Pain/Discomfort: Week 36: number analyzed (Participants) | 395 | 405 | 270 | 177 | 184
  Pain/Discomfort: Week 36: No Problems | 95 | 84 | 55 | 47 | 35
  Pain/Discomfort: Week 36: Slight Problems | 206 | 220 | 127 | 94 | 97
  Pain/Discomfort: Week 36: Moderate Problems | 81 | 89 | 79 | 34 | 45
  Pain/Discomfort: Week 36: Severe Problems | 13 | 11 | 8 | 2 | 7
  Pain/Discomfort: Week 36: Extreme Problems | 0 | 1 | 1 | 0 | 0
  Pain/Discomfort: Week 52: number analyzed (Participants) | 386 | 379 | 257 | 167 | 174
  Pain/Discomfort: Week 52: No Problems | 90 | 88 | 57 | 45 | 44
  Pain/Discomfort: Week 52: Slight Problems | 209 | 210 | 130 | 80 | 93
  Pain/Discomfort: Week 52: Moderate Problems | 77 | 72 | 61 | 38 | 31
  Pain/Discomfort: Week 52: Severe Problems | 10 | 9 | 9 | 3 | 6
  Pain/Discomfort: Week 52: Extreme Problems | 0 | 0 | 0 | 1 | 0
  Anxiety/Depression: Week 36: number analyzed (Participants) | 395 | 405 | 270 | 177 | 184
  Anxiety/Depression: Week 36: No Problems | 230 | 259 | 162 | 115 | 112
  Anxiety/Depression: Week 36: Slight Problems | 123 | 113 | 79 | 44 | 51
  Anxiety/Depression: Week 36: Moderate Problems | 37 | 27 | 19 | 18 | 16
  Anxiety/Depression: Week 36: Severe Problems | 4 | 5 | 7 | 0 | 5
  Anxiety/Depression: Week 36: Extreme Problems | 1 | 1 | 3 | 0 | 0
  Anxiety/Depression: Week 52: number analyzed (Participants) | 386 | 379 | 257 | 167 | 174
  Anxiety/Depression: Week 52: No Problems | 227 | 254 | 169 | 111 | 110
  Anxiety/Depression: Week 52: Slight Problems | 106 | 86 | 61 | 38 | 41
  Anxiety/Depression: Week 52: Moderate Problems | 48 | 34 | 23 | 17 | 19
  Anxiety/Depression: Week 52: Severe Problems | 5 | 5 | 4 | 0 | 4
  Anxiety/Depression: Week 52: Extreme Problems | 0 | 0 | 0 | 1 | 0

61. Secondary Outcome: EQ-5D Current Health VAS at Weeks 4, 12, and 24
Description: EQ-5D-5L is a standardized measure of health status of the participant at the visit (same day) that provides a simple, generic measure of health for clinical and economic appraisal. Participant rates their current health state on a 0-100 VAS. It gets recorded on a vertical VAS in which the endpoints are labeled best imaginable health state is 100 (on the top) and worst imaginable health state is 0 (on the bottom). Higher scores of EQ VAS indicate better health.
Time Frame: Weeks 4, 12, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo
Number analyzed (Participants) | 475 | 480 | 325 | 475
score on a scale
  Week 4: number analyzed (Participants) | 468 | 471 | 319 | 457
  Week 4 | 59 (20.5) | 59 (19.9) | 60 (20.4) | 56 (19.5)
  Week 12: number analyzed (Participants) | 455 | 457 | 307 | 437
  Week 12 | 66 (20.3) | 66 (20.3) | 65 (19.6) | 59 (20.7)
  Week 24: number analyzed (Participants) | 416 | 419 | 277 | 372
  Week 24 | 67 (23.1) | 69 (21.6) | 68 (22.2) | 64 (21.4)

62. Secondary Outcome: EQ-5D Current Health VAS at Weeks 36, and 52
Description: as for outcome 61
Time Frame: Weeks 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Filgotinib 200 mg: Participants were administered a filgotinib 200 mg tablet orally, once daily + a placebo to match (PTM) filgotinib 100 mg tablet orally, once daily + PTM adalimumab 40 mg subcutaneous (SC) injection, once every 2 weeks in addition to a weekly stable dose of MTX, orally median exposure of up to 52.1 weeks.
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo to Filgotinib 200 mg | Placebo to Filgotinib 100 mg
Number analyzed (Participants) | 475 | 480 | 325 | 190 | 191
score on a scale
  Week 36: number analyzed (Participants) | 395 | 405 | 270 | 177 | 184
  Week 36 | 69 (22.7) | 72 (21.2) | 67 (24.3) | 73 (19.9) | 71 (21.1)
  Week 52: number analyzed (Participants) | 386 | 379 | 257 | 167 | 174
  Week 52 | 72 (21.3) | 73 (21.0) | 71 (22.5) | 73 (20.6) | 70 (22.8)

63. Secondary Outcome: Change From Baseline in EQ-5D Current Health VAS at Weeks 4, 12, and 24
Description: The EQ-5D-5L is a standardized measure of health status of the participant at the visit (same day) that provides a simple, generic measure of health for clinical and economic appraisal. Participant rates their current health state on a 0-100 VAS. It gets recorded on a vertical VAS in which the endpoints are labeled best imaginable health state is 100 (on the top) and worst imaginable health state is 0 (on the bottom). Higher scores of EQ VAS indicate better health. Positive change indicates improvement (better health).
Time Frame: Baseline; Weeks 4, 12, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo
Number analyzed (Participants) | 472 | 477 | 319 | 469
score on a scale
  Baseline | 48 (22.5) | 49 (22.8) | 47 (21.8) | 46 (21.8)
  Change from Baseline at Week 4: number analyzed (Participants) | 465 | 470 | 316 | 455
  Change from Baseline at Week 4 | 11 (24.4) | 10 (25.2) | 13 (24.4) | 10 (25.1)
  Change from Baseline at Week 12: number analyzed (Participants) | 452 | 455 | 304 | 432
  Change from Baseline at Week 12 | 18 (26.3) | 17 (27.4) | 17 (27.1) | 13 (26.5)
  Change from Baseline at Week 24: number analyzed (Participants) | 413 | 417 | 273 | 369
  Change from Baseline at Week 24 | 19 (30.5) | 21 (28.9) | 21 (28.8) | 18 (29.3)
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 14, analysis 3]; Test type: Superiority; p = 0.049, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 2.0, 95% CI 2-sided [0.0 to 5.0], Standard Error of Mean 1.2
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 14, analysis 4]; Test type: Superiority; p = 0.069, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 2.0, 95% CI 2-sided [-0.0 to 5.0], Standard Error of Mean 1.2
Statistical Analysis 3: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 7.0, 95% CI 2-sided [4.0 to 9.0], Standard Error of Mean 1.3
Statistical Analysis 4: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 6.0, 95% CI 2-sided [4.0 to 9.0], Standard Error of Mean 1.3
Statistical Analysis 5: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.060, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 3.0, 95% CI 2-sided [-0.0 to 6.0], Standard Error of Mean 1.5
Statistical Analysis 6: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p = 0.003, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 5.0, 95% CI 2-sided [2.0 to 8.0], Standard Error of Mean 1.5

64. Secondary Outcome: Change From Baseline in EQ-5D Current Health VAS at Weeks 36, and 52
Description: as for outcome 63
Time Frame: Baseline; Weeks 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo to Filgotinib 200 mg | Placebo to Filgotinib 100 mg
Number analyzed (Participants) | 472 | 477 | 319 | 189 | 189
score on a scale
  Baseline | 48 (22.5) | 49 (22.8) | 47 (21.8) | 45 (21.6) | 47 (21.1)
  Change from Baseline at Week 36: number analyzed (Participants) | 393 | 403 | 268 | 176 | 182
  Change from Baseline at Week 36 | 21 (30.6) | 23 (28.5) | 20 (30.9) | 28 (28.2) | 24 (26.0)
  Change from Baseline at Week 52: number analyzed (Participants) | 384 | 376 | 254 | 166 | 172
  Change from Baseline at Week 52 | 25 (29.3) | 24 (28.5) | 24 (29.2) | 29 (28.6) | 23 (29.6)

65. Secondary Outcome: Work Productivity and Activity Impairment-Rheumatoid Arthritis (WPAI-RA): Mean Percentage of Work Time Missed (Absenteeism) at Weeks 4, 12, and 24
Description: The WPAI is a questionnaire that measures impairments in work activities in participants with RA which consists of 6 questions: Q1-currently employed; Q2-work time missed due to RA; Q3-work time missed due to other reasons; Q4-hours actually worked; Q5-degree RA affected productivity while working (0-10 VAS, with 0 indicating no effect and 10 indicating RA completely prevented the participant from working); Q6-degree RA affected productivity in regular unpaid activities (0-10 VAS, with 0 indicating no effect and 10 indicating RA completely prevented the participant's daily activities). Outcomes are expressed as impairment percentages: Absenteeism (work time missed) due to RA: 100×{Q2/(Q2+Q4)}. Higher numbers indicate greater impairment and less productivity.
Time Frame: Weeks 4, 12, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of work time missed
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo
Number analyzed (Participants) | 475 | 480 | 325 | 475
percentage of work time missed
  Week 4: number analyzed (Participants) | 191 | 185 | 112 | 161
  Week 4 | 8.5 (21.27) | 6.6 (16.47) | 9.2 (21.99) | 9.4 (21.41)
  Week 12: number analyzed (Participants) | 189 | 177 | 111 | 153
  Week 12 | 6.6 (17.06) | 5.4 (14.56) | 7.1 (18.46) | 9.5 (22.66)
  Week 24: number analyzed (Participants) | 178 | 168 | 112 | 132
  Week 24 | 4.4 (13.54) | 3.6 (10.24) | 7.2 (17.72) | 10.5 (21.86)

66. Secondary Outcome: WPAI-RA: Mean Percentage of Work Time Missed (Absenteeism) at Weeks 36, and 52
Description: as for outcome 65
Time Frame: Weeks 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of work time missed
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo to Filgotinib 200 mg | Placebo to Filgotinib 100 mg
Number analyzed (Participants) | 475 | 480 | 325 | 190 | 191
percentage of work time missed
  Week 36: number analyzed (Participants) | 178 | 169 | 106 | 72 | 63
  Week 36 | 5.5 (16.17) | 7.7 (19.46) | 7.0 (19.65) | 6.8 (19.79) | 8.4 (19.97)
  Week 52: number analyzed (Participants) | 180 | 156 | 99 | 66 | 55
  Week 52 | 4.8 (14.39) | 5.4 (15.10) | 7.4 (20.12) | 5.5 (13.24) | 5.8 (14.29)

67. Secondary Outcome: WPAI-RA: Mean Percentage of Impairment While Working Due to RA (Presenteeism) at Weeks 4, 12, and 24
Description: The WPAI is a questionnaire that measures impairments in work activities in participants with RA which consists of 6 questions: Q1-currently employed; Q2-work time missed due to RA; Q3-work time missed due to other reasons; Q4-hours actually worked; Q5-degree RA affected productivity while working (0-10 VAS, with 0 indicating no effect and 10 indicating RA completely prevented the participant from working); Q6-degree RA affected productivity in regular unpaid activities (0-10 VAS, with 0 indicating no effect and 10 indicating RA completely prevented the participant's daily activities). Outcomes are expressed as impairment percentages: Presenteeism (impairment while working) due to RA: 100×{Q5/10}. Higher numbers indicate greater impairment and less productivity.
Time Frame: Weeks 4, 12, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of impairment while working
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo
Number analyzed (Participants) | 475 | 480 | 325 | 475
percentage of impairment while working
  Week 4: number analyzed (Participants) | 185 | 182 | 108 | 156
  Week 4 | 34.3 (22.69) | 36.9 (24.01) | 35.6 (22.39) | 42.5 (23.54)
  Week 12: number analyzed (Participants) | 187 | 176 | 109 | 147
  Week 12 | 26.3 (21.07) | 26.9 (22.57) | 27.6 (21.51) | 34.0 (21.98)
  Week 24: number analyzed (Participants) | 177 | 168 | 110 | 128
  Week 24 | 22.0 (21.28) | 21.0 (20.74) | 25.7 (21.99) | 30.9 (23.11)

68. Secondary Outcome: WPAI-RA: Mean Percentage of Impairment While Working Due to RA (Presenteeism) at Weeks 36, and 52
Description: as for outcome 67
Time Frame: Weeks 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of impairment while working
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo to Filgotinib 200 mg | Placebo to Filgotinib 100 mg
Number analyzed (Participants) | 475 | 480 | 325 | 190 | 191
percentage of impairment while working
  Week 36: number analyzed (Participants) | 176 | 166 | 103 | 71 | 62
  Week 36 | 20.2 (19.54) | 19.6 (20.27) | 21.2 (20.74) | 21.5 (18.72) | 25.8 (23.51)
  Week 52: number analyzed (Participants) | 179 | 155 | 97 | 66 | 55
  Week 52 | 18.2 (18.83) | 17.3 (19.25) | 20.8 (21.78) | 22.3 (21.82) | 19.5 (20.04)

69. Secondary Outcome: WPAI-RA: Mean Percentage of Overall Work Productivity Impairment Due to RA at Weeks 4, 12, and 24
Description: The WPAI is a questionnaire that measures impairments in work activities in participants with RA which consists of 6 questions: Q1-currently employed; Q2-work time missed due to RA; Q3-work time missed due to other reasons; Q4-hours actually worked; Q5-degree RA affected productivity while working (0-10 VAS, with 0 indicating no effect and 10 indicating RA completely prevented the participant from working); Q6-degree RA affected productivity in regular unpaid activities (0-10 VAS, with 0 indicating no effect and 10 indicating RA completely prevented the participant's daily activities). Outcomes are expressed as impairment percentages: Work productivity loss (overall work impairment) due to RA: 100×{Q2/(Q2+Q4) + [(1-Q2/(Q2+Q4) × (Q5/10)]}. Higher numbers indicate greater impairment and less productivity.
Time Frame: Weeks 4, 12, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of work productivity loss
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo
Number analyzed (Participants) | 475 | 480 | 325 | 475
percentage of work productivity loss
  Week 4: number analyzed (Participants) | 185 | 182 | 108 | 156
  Week 4 | 37.0 (24.64) | 39.5 (25.17) | 38.4 (24.59) | 45.1 (25.18)
  Week 12: number analyzed (Participants) | 187 | 176 | 109 | 147
  Week 12 | 29.5 (24.25) | 29.3 (24.73) | 30.7 (24.34) | 36.7 (24.27)
  Week 24: number analyzed (Participants) | 177 | 168 | 110 | 128
  Week 24 | 24.4 (23.06) | 23.2 (22.64) | 29.1 (23.88) | 34.9 (26.04)

70. Secondary Outcome: WPAI-RA: Mean Percentage of Overall Work Productivity Impairment Due to RA at Weeks 36, and 52
Description: as for outcome 69
Time Frame: Weeks 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of work productivity loss
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo to Filgotinib 200 mg | Placebo to Filgotinib 100 mg
Number analyzed (Participants) | 475 | 480 | 325 | 190 | 191
percentage of work productivity loss
  Week 36: number analyzed (Participants) | 176 | 166 | 103 | 71 | 62
  Week 36 | 23.3 (22.02) | 23.9 (23.98) | 23.8 (22.95) | 24.0 (21.33) | 29.1 (26.79)
  Week 52: number analyzed (Participants) | 179 | 155 | 97 | 66 | 55
  Week 52 | 20.6 (21.74) | 20.5 (22.15) | 24.3 (24.77) | 25.7 (24.32) | 22.3 (24.10)

71. Secondary Outcome: WPAI-RA: Mean Percentage of Activity Impairment Due to RA at Weeks 4, 12, and 24
Description: The WPAI is a questionnaire that measures impairments in work activities in participants with RA which consists of 6 questions: Q1-currently employed; Q2-work time missed due to RA; Q3-work time missed due to other reasons; Q4-hours actually worked; Q5-degree RA affected productivity while working (0-10 VAS, with 0 indicating no effect and 10 indicating RA completely prevented the participant from working); Q6-degree RA affected productivity in regular unpaid activities (0-10 VAS, with 0 indicating no effect and 10 indicating RA completely prevented the participant's daily activities). Outcomes are expressed as impairment percentages: Activity impairment due to RA: 100×{Q6/10}. If Question 1 (Are you currently employed?) is 'NO', then only the activity impairment score can be determined. Higher numbers indicate greater impairment and less productivity.
Time Frame: Weeks 4, 12, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of activity impairment
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo
Number analyzed (Participants) | 475 | 480 | 325 | 475
percentage of activity impairment
  Week 4: number analyzed (Participants) | 468 | 471 | 319 | 457
  Week 4 | 44.6 (24.18) | 46.2 (24.05) | 46.4 (23.84) | 52.1 (23.41)
  Week 12: number analyzed (Participants) | 455 | 457 | 306 | 437
  Week 12 | 35.1 (23.86) | 36.6 (24.51) | 38.3 (25.57) | 44.3 (23.73)
  Week 24: number analyzed (Participants) | 416 | 419 | 277 | 372
  Week 24 | 30.2 (24.69) | 30.4 (23.07) | 32.5 (24.40) | 39.3 (23.69)

72. Secondary Outcome: WPAI-RA: Mean Percentage of Activity Impairment Due to RA at Weeks 36, and 52
Description: as for outcome 71
Time Frame: Weeks 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of activity impairment
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo to Filgotinib 200 mg | Placebo to Filgotinib 100 mg
Number analyzed (Participants) | 475 | 480 | 325 | 190 | 191
percentage of activity impairment
  Week 36: number analyzed (Participants) | 395 | 404 | 270 | 177 | 184
  Week 36 | 28.3 (23.30) | 28.7 (23.47) | 31.3 (25.44) | 28.3 (22.47) | 32.3 (23.62)
  Week 52: number analyzed (Participants) | 386 | 379 | 257 | 167 | 174
  Week 52 | 26.0 (22.44) | 26.3 (22.71) | 28.1 (24.38) | 28.6 (23.57) | 28.9 (23.07)

73. Secondary Outcome: Change From Baseline in WPAI-RA: Mean Percentage of Work Time Missed (Absenteeism) at Weeks 4, 12, and 24
Description: The WPAI is a questionnaire that measures impairments in work activities in participants with RA which consists of 6 questions: Q1-currently employed; Q2-work time missed due to RA; Q3-work time missed due to other reasons; Q4-hours actually worked; Q5-degree RA affected productivity while working (0-10 VAS, with 0 indicating no effect and 10 indicating RA completely prevented the participant from working); Q6-degree RA affected productivity in regular unpaid activities (0-10 VAS, with 0 indicating no effect and 10 indicating RA completely prevented the participant's daily activities). Outcomes are expressed as impairment percentages: Absenteeism (work time missed) due to RA: 100×{Q2/(Q2+Q4)}. Higher numbers indicate greater impairment and less productivity. A negative change from baseline indicates improvement.
Time Frame: Baseline; Weeks 4, 12, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of work time missed
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo
Number analyzed (Participants) | 195 | 193 | 127 | 162
percentage of work time missed
  Baseline | 12.0 (25.77) | 9.9 (20.91) | 16.0 (27.57) | 17.0 (29.52)
  Change from Baseline at Week 4: number analyzed (Participants) | 176 | 169 | 107 | 143
  Change from Baseline at Week 4 | -1.4 (21.24) | -2.1 (18.14) | -7.5 (24.26) | -5.7 (25.65)
  Change from Baseline at Week 12: number analyzed (Participants) | 167 | 160 | 103 | 129
  Change from Baseline at Week 12 | -4.3 (22.55) | -3.8 (18.37) | -7.5 (28.79) | -5.9 (27.94)
  Change from Baseline at Week 24: number analyzed (Participants) | 157 | 148 | 100 | 110
  Change from Baseline at Week 24 | -6.1 (24.77) | -3.8 (16.92) | -9.3 (28.99) | -1.5 (27.24)

74. Secondary Outcome: Change From Baseline in WPAI-RA: Mean Percentage of Work Time Missed (Absenteeism) at Weeks 36, and 52
Description: as for outcome 73
Time Frame: Baseline; Weeks 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of work time missed
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo to Filgotinib 200 mg | Placebo to Filgotinib 100 mg
Number analyzed (Participants) | 195 | 193 | 127 | 76 | 62
percentage of work time missed
  Baseline | 12.0 (25.77) | 9.9 (20.91) | 16.0 (27.57) | 18.3 (31.61) | 14.6 (26.88)
  Change from Baseline at Week 36: number analyzed (Participants) | 149 | 143 | 94 | 63 | 48
  Change from Baseline at Week 36 | -4.4 (24.04) | -1.5 (24.41) | -8.7 (27.43) | -6.2 (30.25) | -7.5 (25.00)
  Change from Baseline at Week 52: number analyzed (Participants) | 154 | 131 | 89 | 55 | 43
  Change from Baseline at Week 52 | -6.8 (26.27) | -1.7 (21.89) | -7.1 (24.00) | -7.4 (26.76) | -8.9 (27.90)

75. Secondary Outcome: Change From Baseline in WPAI-RA: Mean Percentage of Impairment While Working Due to RA (Presenteeism) at Weeks 4, 12, and 24
Description: The WPAI is a questionnaire that measures impairments in work activities in participants with RA which consists of 6 questions: Q1-currently employed; Q2-work time missed due to RA; Q3-work time missed due to other reasons; Q4-hours actually worked; Q5-degree RA affected productivity while working (0-10 VAS, with 0 indicating no effect and 10 indicating RA completely prevented the participant from working); Q6-degree RA affected productivity in regular unpaid activities (0-10 VAS, with 0 indicating no effect and 10 indicating RA completely prevented the participant's daily activities). Outcomes are expressed as impairment percentages: Presenteeism (impairment while working) due to RA: 100×{Q5/10}. Higher numbers indicate greater impairment and less productivity. A negative change from baseline indicates improvement.
Time Frame: Baseline; Weeks 4, 12, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of impairment while working
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo
Number analyzed (Participants) | 184 | 187 | 119 | 150
percentage of impairment while working
  Baseline | 49.1 (25.23) | 48.0 (24.61) | 50.8 (22.98) | 52.5 (25.89)
  Change from Baseline at Week 4: number analyzed (Participants) | 166 | 164 | 100 | 132
  Change from Baseline at Week 4 | -15.1 (23.19) | -10.2 (22.82) | -15.3 (24.84) | -9.5 (23.68)
  Change from Baseline at Week 12: number analyzed (Participants) | 160 | 156 | 96 | 118
  Change from Baseline at Week 12 | -24.1 (25.83) | -21.9 (23.22) | -22.9 (24.88) | -17.1 (27.24)
  Change from Baseline at Week 24: number analyzed (Participants) | 151 | 146 | 93 | 102
  Change from Baseline at Week 24 | -27.4 (26.37) | -25.9 (26.59) | -23.3 (27.56) | -21.2 (29.33)

76. Secondary Outcome: Change From Baseline in WPAI-RA: Mean Percentage of Impairment While Working Due to RA (Presenteeism) at Weeks 36, and 52
Description: as for outcome 75
Time Frame: Baseline; Weeks 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of impairment while working
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo to Filgotinib 200 mg | Placebo to Filgotinib 100 mg
Number analyzed (Participants) | 184 | 187 | 119 | 69 | 59
percentage of impairment while working
  Baseline | 49.1 (25.23) | 48.0 (24.61) | 50.8 (22.98) | 53.8 (26.35) | 53.6 (23.40)
  Change from Baseline at Week 36: number analyzed (Participants) | 144 | 138 | 87 | 61 | 45
  Change from Baseline at Week 36 | -29.7 (26.73) | -27.5 (26.28) | -27.8 (29.90) | -32.0 (26.82) | -26.4 (29.86)
  Change from Baseline at Week 52: number analyzed (Participants) | 144 | 128 | 84 | 52 | 40
  Change from Baseline at Week 52 | -31.7 (27.44) | -29.5 (24.66) | -29.4 (27.91) | -30.6 (28.24) | -32.5 (28.17)

77. Secondary Outcome: Change From Baseline in WPAI-RA: Mean Percentage of Overall Work Productivity Impairment Due to RA at Weeks 4, 12, and 24
Description: The WPAI is a questionnaire that measures impairments in work activities in participants with RA which consists of 6 questions: Q1-currently employed; Q2-work time missed due to RA; Q3-work time missed due to other reasons; Q4-hours actually worked; Q5-degree RA affected productivity while working (0-10 VAS, with 0 indicating no effect and 10 indicating RA completely prevented the participant from working); Q6-degree RA affected productivity in regular unpaid activities (0-10 VAS, with 0 indicating no effect and 10 indicating RA completely prevented the participant's daily activities). Outcomes are expressed as impairment percentages: Work productivity loss (overall work impairment) due to RA: 100×{Q2/(Q2+Q4) + [(1-Q2/(Q2+Q4) × (Q5/10)]}. Higher numbers indicate greater impairment and less productivity. A negative change from baseline indicates improvement.
Time Frame: Baseline; Weeks 4, 12, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of work productivity loss
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo
Number analyzed (Participants) | 184 | 187 | 119 | 150
percentage of work productivity loss
  Baseline | 51.3 (25.95) | 50.6 (25.87) | 54.3 (24.85) | 55.8 (27.33)
  Change from Baseline at Week 4: number analyzed (Participants) | 166 | 164 | 100 | 132
  Change from Baseline at Week 4 | -14.6 (24.59) | -10.2 (23.71) | -16.8 (26.29) | -10.0 (24.06)
  Change from Baseline at Week 12: number analyzed (Participants) | 160 | 156 | 96 | 118
  Change from Baseline at Week 12 | -23.2 (28.18) | -22.3 (24.34) | -22.8 (26.61) | -17.5 (28.09)
  Change from Baseline at Week 24: number analyzed (Participants) | 151 | 146 | 93 | 102
  Change from Baseline at Week 24 | -27.1 (27.78) | -26.3 (27.29) | -23.6 (29.40) | -19.3 (30.81)

78. Secondary Outcome: Change From Baseline in WPAI-RA: Mean Percentage of Overall Work Productivity Impairment Due to RA at Weeks 36, and 52
Description: as for outcome 77
Time Frame: Baseline; Weeks 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of work productivity loss
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo to Filgotinib 200 mg | Placebo to Filgotinib 100 mg
Number analyzed (Participants) | 184 | 187 | 119 | 69 | 59
percentage of work productivity loss
  Baseline | 51.3 (25.95) | 50.6 (25.87) | 54.3 (24.85) | 56.6 (27.36) | 57.1 (25.14)
  Change from Baseline at Week 36: number analyzed (Participants) | 144 | 138 | 87 | 61 | 45
  Change from Baseline at Week 36 | -28.9 (27.16) | -25.7 (29.54) | -28.6 (31.48) | -31.7 (30.53) | -26.9 (31.02)
  Change from Baseline at Week 52: number analyzed (Participants) | 144 | 128 | 84 | 52 | 40
  Change from Baseline at Week 52 | -31.6 (29.17) | -28.4 (27.11) | -29.3 (29.38) | -30.3 (30.73) | -32.7 (29.65)

79. Secondary Outcome: Change From Baseline in WPAI-RA: Mean Percentage of Activity Impairment Due to RA at Weeks 4, 12, and 24
Description: The WPAI is a questionnaire that measures impairments in work activities in participants with RA which consists of 6 questions: Q1-currently employed; Q2-work time missed due to RA; Q3-work time missed due to other reasons; Q4-hours actually worked; Q5-degree RA affected productivity while working (0-10 VAS, with 0 indicating no effect and 10 indicating RA completely prevented the participant from working); Q6-degree RA affected productivity in regular unpaid activities (0-10 VAS, with 0 indicating no effect and 10 indicating RA completely prevented the participant's daily activities). Outcomes are expressed as impairment percentages: Activity impairment due to RA: 100×{Q6/10}. If Question 1 (Are you currently employed?) is 'NO', then only the activity impairment score can be determined. Higher numbers indicate greater impairment and less productivity. A negative change from baseline indicates improvement.
Time Frame: Baseline; Weeks 4, 12, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of activity impairment
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo
Number analyzed (Participants) | 472 | 477 | 319 | 469
percentage of activity impairment
  Baseline | 61.5 (22.74) | 60.5 (23.85) | 61.3 (21.20) | 62.2 (22.11)
  Change from Baseline at Week 4: number analyzed (Participants) | 465 | 470 | 316 | 455
  Change from Baseline at Week 4 | -17.0 (22.46) | -14.7 (22.07) | -14.8 (23.36) | -9.8 (20.98)
  Change from Baseline at Week 12: number analyzed (Participants) | 452 | 455 | 303 | 432
  Change from Baseline at Week 12 | -26.5 (25.17) | -24.1 (24.95) | -22.6 (24.93) | -16.9 (25.98)
  Change from Baseline at Week 24: number analyzed (Participants) | 413 | 417 | 273 | 369
  Change from Baseline at Week 24 | -30.7 (26.20) | -30.4 (25.45) | -28.6 (24.99) | -21.9 (27.78)

80. Secondary Outcome: Change From Baseline in WPAI-RA: Mean Percentage of Activity Impairment Due to RA at Weeks 36, and 52
Description: as for outcome 79
Time Frame: Baseline; Weeks 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of activity impairment
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo to Filgotinib 200 mg | Placebo to Filgotinib 100 mg
Number analyzed (Participants) | 472 | 477 | 319 | 189 | 189
percentage of activity impairment
  Baseline | 61.5 (22.74) | 60.5 (23.85) | 61.3 (21.20) | 62.9 (21.74) | 59.7 (22.10)
  Change from Baseline at Week 36: number analyzed (Participants) | 393 | 402 | 268 | 176 | 182
  Change from Baseline at Week 36 | -32.6 (26.66) | -31.5 (25.66) | -30.2 (26.93) | -34.9 (26.60) | -27.5 (26.14)
  Change from Baseline at Week 52: number analyzed (Participants) | 384 | 376 | 254 | 166 | 172
  Change from Baseline at Week 52 | -34.8 (26.74) | -33.7 (26.44) | -32.9 (26.03) | -35.2 (28.00) | -30.8 (25.99)

ADVERSE EVENTS:
Time Frame: First dose date up to last dose date (Maximum: 54 weeks) plus 30 days
Description: The Safety Analysis Set included all participants who received at least 1 dose of study drug.
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Adalimumab | Placebo to Filgotinib 200 mg | Placebo to Filgotinib 100 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 3/475 | 1/480 | 1/325 | 1/190 | 1/191 | 2/475
Serious Adverse Events (participants affected / at risk) | 35/475 | 40/480 | 22/325 | 7/190 | 8/191 | 21/475
Other Adverse Events (participants affected / at risk) | 128/475 | 142/480 | 82/325 | 36/190 | 23/191 | 61/475
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Filgotinib 200 mg (N=475) | Filgotinib 100 mg (N=480) | Adalimumab (N=325) | Placebo to Filgotinib 200 mg (N=190) | Placebo to Filgotinib 100 mg (N=191) | Placebo (N=475)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1
Angina unstable (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cor pulmonale chronic (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Meniere's disease (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 1
Macular fibrosis (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vitreous opacities (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 1 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Obstructive pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Peptic ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 1 | 0 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Arthritis infective (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 1
Candida infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Helicobacter infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Infected skin ulcer (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Infectious pleural effusion (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Infective tenosynovitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 4 | 4 | 3 | 1 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
Pneumonia fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia pneumococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Septic shock (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Varicella (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Coronary artery restenosis (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypervitaminosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0
Limb asymmetry (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Cervix carcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Leiomyosarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Malignant glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Hemiplegia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Prerenal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Renal cell dysplasia (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rheumatoid lung (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Peripheral artery occlusion (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Filgotinib 200 mg (N=475) | Filgotinib 100 mg (N=480) | Adalimumab (N=325) | Placebo to Filgotinib 200 mg (N=190) | Placebo to Filgotinib 100 mg (N=191) | Placebo (N=475)
Nausea (Gastrointestinal disorders) | 26 | 16 | 6 | 4 | 1 | 7
Nasopharyngitis (Infections and infestations) | 43 | 48 | 24 | 7 | 6 | 25
Upper respiratory tract infection (Infections and infestations) | 41 | 49 | 21 | 8 | 6 | 14
Urinary tract infection (Infections and infestations) | 18 | 19 | 17 | 10 | 8 | 6
Alanine aminotransferase increased (Investigations) | 17 | 25 | 21 | 7 | 3 | 11
Aspartate aminotransferase increased (Investigations) | 12 | 20 | 17 | 8 | 3 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2016-07-05): https://cdn.clinicaltrials.gov/large-docs/96/NCT02889796/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-05): https://cdn.clinicaltrials.gov/large-docs/96/NCT02889796/SAP_001.pdf